CLINICAL TRIAL: NCT01597635
Title: A Two Part Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK2586881 in Patients With Acute Lung Injury
Brief Title: The Safety, Tolerability, PK and PD of GSK2586881 in Patients With Acute Lung Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 114622
Record Dates: First submitted 2012-01-26; First posted 2012-05-14 (Estimated); Results first posted 2017-09-28 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-08

CONDITIONS: Lung Injury, Acute
Keywords: rhACE2; Acute Respiratory Distress Syndrome (ARDS); Acute Lung Injury; GSK2586881; critical care
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): 4 increasing doses of GSK2586881 given over 2 days
  Interventions: Drug: Dose 1 GSK2586881; Drug: Dose 2 GSK2586881; Drug: Dose 3 GSK2586881; Drug: Dose 4 GSK2586881
- Part B (Experimental): Repeat Medium-High dose of GSK2586881 (or placebo) over 3 days
  Interventions: Drug: Dose 3 GSK2586881; Drug: Placebo (saline)

INTERVENTIONS:
Drug: Dose 1 GSK2586881 — Low dose GSK2586881 administered intravenously
  Arms: Part A
Drug: Dose 2 GSK2586881 — Medium dose GSK2586881 administered intravenously
  Arms: Part A
Drug: Dose 3 GSK2586881 — Medium-High dose GSK2586881 administered intravenously
Drug: Dose 4 GSK2586881 — High dose GSK2586881 administered intravenously
  Arms: Part A
Drug: Placebo (saline) — Administered intravenously to match intervention
  Arms: Part B

SUMMARY:
This is an early phase (phase IIa), randomized, multi-center study in subjects with acute lung injury (ALI) or acute respiratory distress syndrome (ARDS). The purpose of this study is to investigate the safety of GSK2586881 and to determine what effects it has on people with Acute Lung Injury (ALI) or Acute Respiratory Distress Syndrome (ARDS).

The study has two parts: Part A will be an open-label investigation in five subjects. Part B will be a double-blind, placebo controlled investigation and will involve approximately 60 subjects.

DETAILED DESCRIPTION:
The acute respiratory distress syndrome (ARDS) is a form of severe acute lung injury (ALI) characterized by hypoxemic respiratory failure (the lungs are unable to absorb oxygen to the arterial blood) and non-cardiogenic pulmonary edema (accumulation of fluid in the lungs). The syndrome may be caused by direct or indirect injury to the lungs. It is associated with a mortality rate of up to 40-50%. There are no marketed pharmacologic therapies for this devastating syndrome.

This study aims to assess the safety, tolerability and pharmacodynamics of GSK2586881, a recombinant human angiotensin converting enzyme type 2 (rhACE2).

ACE2 is involved in the Renin-Angiotensin System (RAS), which controls blood pressure, electrolytes and intravascular fluid volume. A key function of rhACE2 is believed to be the cleavage of Angiotensin II (Ang II) to Ang (1-7), which have opposing physiological roles. Elevated levels of Ang II are associated with vasoconstriction, inflammation, fibrosis, vascular leak, and sodium absorption. Ang (1-7) appears to be a counterregulatory protein in the RAS; associated with vasodilation, anti-proliferation, antiinflammation, and reduced vascular leak. It has been observed that levels of Ang II are increased in humans with ALI/ ARDS. It is expected that the reduction of Ang II should have a positive impact on ALI and ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 - 80 years of age (inclusive)
* Diagnosis of ALI with acute onset of PaO2/FiO2 ratio less than or equal to 300, and bilateral infiltrates consistent with pulmonary edema on frontal chest radiograph. The infiltrates may be patchy, diffuse, homogeneous, or asymmetric, and requirement for positive pressure ventilation via an endotracheal tube, and no clinical evidence of left atrial hypertension
* Cause of ALI thought to be associated with infection, sepsis, pneumonia, aspiration, or similar as judged by the PI and/or medical monitor
* The subject must be randomized into the study within 48 hours from the time of diagnosis of ALI
* Period of hemodynamic stability (e.g. 4-6 hours) prior to the initiation of study treatment not requiring resuscitative measures with stable pressor requirements. In this study low-dose arginine vasopressin is not considered a pressor, and is permitted in Parts A and B.
* If mechanically ventilated, duration of mechanical ventilation must be less than 72 hours before dosing begins
* BMI within the range 19.0 - 38.0 kg/m2 inclusive
* The subject or legal decision maker is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB or QTcF less than 450 msec; or QTc less than 480 msec in subjects with Bundle Branch Block.
* Alanine aminotransferase (ALT) less than 5 x Upper Limit of Normal (ULN); bilirubin less than or equal to 1.5 x ULN.

Exclusion Criteria:

* Subjects whose clinical condition is deteriorating rapidly or any subject for whom the investigator does not consider there is a reasonable expectation that they will be able to complete the study.
* Known positive Hepatitis B surface antigen, Hepatitis C antibody or HIV antibody
* Current or chronic history of liver disease (Child Pugh score of greater than or equal to 10), or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Known history of substance abuse or alcohol abuse, within 6 months of the study causing chronic liver disease such as cirrhosis, chronic ascites or portal hypertension, or known evidence of withdrawal syndrome within the past 6 months.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Inability to discontinue use of Angiotensin converting enzyme type 1 inhibitors or Angiotensin receptor blockers.
* Patients requiring high doses of loop diuretics with significant intravascular volume depletion, as assessed clinically
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* Pregnant females as determined by positive serum or urine hCG test prior to dosing
* Lactating females
* Unwillingness or inability to follow the procedures outlined in the protocol
* Subject is legally incapacitated (e.g. a prisoner)
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* Unstable Hemoglobin (Hb less than 7) at time of drug infusion
* Malignancy or other irreversible condition for which 6 month mortality is estimated to be greater than 50%
* Arterial blood pH less than 7.1 or serum HCO3 - less than 15 (if ABG not available) before infusion is started
* Known severe chronic respiratory disease:
* known Forced Expiratory Volume in 1 second (FEV1)/ Forced Vital Capacity (FVC) less than 45% predicted, or
* known chronic hypercapnia (PaCO2 greater than 45 mmHg) or chronic hypoxemia (PaO2 less than 55 mmHg) on FiO2 =0.21, or
* known FEV1 less than 15 ml/kg (e.g. 1L for 70 kg person), or
* known radiographic evidence of chronic interstitial infiltration, or
* known hospitalization within the past six months for respiratory failure (PaCO2 greater than 50 mmHg or PaO2 less than 55 mmHg, or oxygen saturation less than 88% on FiO2 = 0.21), or
* known chronic restrictive, obstructive, neuromuscular, chest wall, or pulmonary vascular disease resulting in severe exercise restriction
* Known history of neuromuscular disease that would affect time on mechanical ventilation or impairs ability to ventilate spontaneously
* Vasculitis with diffuse alveolar hemorrhage
* Lung transplantation
* Pre-existing renal failure on hemodialysis or peritoneal dialysis requiring renal replacement therapy
* A patient will be excluded if in the judgement of the Principle Investigator or GSK medical monitor their participation could jeopardize the health of the subject or the integrity of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-09-01; Primary Completion 2014-10-01 (Actual); Study Completion 2014-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- United States (12):
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
- Canada (5):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec

REFERENCES:
- [Derived] Khan A, Benthin C, Zeno B, Albertson TE, Boyd J, Christie JD, Hall R, Poirier G, Ronco JJ, Tidswell M, Hardes K, Powley WM, Wright TJ, Siederer SK, Fairman DA, Lipson DA, Bayliffe AI, Lazaar AL. A pilot clinical trial of recombinant human angiotensin-converting enzyme 2 in acute respiratory distress syndrome. Crit Care. 2017 Sep 7;21(1):234. doi: 10.1186/s13054-017-1823-x. PMID 28877748

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted across 5 centers in United States and 5 centers in Canada from 20 September 2012 to 06 October 2014.
Pre-assignment Details: A total of 46 participants were randomized for this study of which 44 participants (5 participants in Part A and 39 participants in Part B) received at least one dose of study medication.
Groups:
- Part A: Eligible participants received multiple single intravenous escalating doses of GSK2586881 (0.1 milligrams per kilograms [mg/kg], 0.2 mg/kg, 0.4 mg/kg, 0.8 mg/kg) as a slow infusion over 3-5 minutes over 2 days.
- Part B (Placebo BID): Eligible participants received intravenous matching placebo (saline solution) twice daily (BID) as a slow infusion over 3-5 minutes for 3 days.
- Part B (GSK2586881 BID): Eligible participants received intravenous dose of 0.4 mg/kg BID of GSK2586881 as a slow infusion over 3-5 minutes for 3 days.
Period: Part A
Arm/Group | Part A | Part B (Placebo BID) | Part B (GSK2586881 BID)
Started | 5 | 0 | 0
Completed | 2 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0
Period: Part B
Arm/Group | Part A | Part B (Placebo BID) | Part B (GSK2586881 BID)
Started | 0 | 20 | 19
Completed | 0 | 14 | 15
Not Completed | 0 | 6 | 4
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Protocol-defined stopping criteria | 0 | 4 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A: Eligible participants received multiple single intravenous escalating doses of GSK2586881 (0.1 mg/kg, 0.2 mg/kg, 0.4 mg/kg, 0.8 mg/kg) as a slow infusion over 3-5 minutes over 2 days.
- Part B (Placebo BID): Eligible participants received intravenous matching placebo (saline solution) BID as a slow infusion over 3-5 minutes for 3 days.
- Total: Total of all reporting groups
Arm/Group | Part A | Part B (Placebo BID) | Part B (GSK2586881 BID) | Total
Number analyzed (Participants) | 5 | 20 | 19 | 44
Age, Customized [Count of Participants; unit: Participants]
  18-80 years | 5 | 20 | 19 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 6 | 15
  Male | 3 | 13 | 13 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 5 | 17 | 18 | 40
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate Assessments Upto Day 7 (Part B)
Description: Vital sign included heart rate. Assessments were performed at Pre-dose, 0.5 hours, 2 hours, 6 hours and 12 hours on Day 1, 0 hours on Day 2 at 0 hours, 0.5 hours, 2 hours, 6 hours, 12 hours, 18 hours and 24 hours on Day 3 and at follow-up on Day 7.
Time Frame: Up to Day 7
Population: The All Subjects - Part B Population was defined as all participants in Part B who received at least one dose of study medication. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
Beats per minute
  Heart rate on Day 1 at Pre-dose | 87.4 (16.32) | 97.7 (16.25)
  Heart rate on Day 1 at 0.5 hours | 87.9 (17.08) | 95.3 (15.10)
  Heart rate on Day 1 at 2 hours | 88.8 (18.22) | 94.7 (17.59)
  Heart rate on Day 1 at 6 hours | 90.0 (18.03) | 96.5 (18.58)
  Heart rate on Day 1 at 12 hours | 87.6 (20.60) | 97.1 (18.46)
  Heart rate on Day 2 at 0 hours | 92.2 (19.02) | 93.4 (16.98)
  Heart rate on Day 3 at 0 hours: number analyzed (Participants) | 18 | 19
  Heart rate on Day 3 at 0 hours | 93.3 (19.20) | 97.7 (14.11)
  Heart rate on Day 3 at 0.5 hours: number analyzed (Participants) | 18 | 19
  Heart rate on Day 3 at 0.5 hours | 91.7 (16.29) | 97.2 (12.81)
  Heart rate on Day 3 at 2 hours: number analyzed (Participants) | 18 | 19
  Heart rate on Day 3 at 2 hours | 93.2 (16.51) | 95.2 (13.31)
  Heart rate on Day 3 at 6 hours: number analyzed (Participants) | 18 | 19
  Heart rate on Day 3 at 6 hours | 93.2 (16.63) | 97.5 (14.44)
  Heart rate on Day 3 at 12 hours: number analyzed (Participants) | 18 | 19
  Heart rate on Day 3 at 12 hours | 93.8 (20.12) | 93.6 (16.08)
  Heart rate on Day 3 at 18 hours: number analyzed (Participants) | 17 | 17
  Heart rate on Day 3 at 18 hours | 98.1 (19.34) | 88.9 (15.69)
  Heart rate on Day 3 at 24 hours: number analyzed (Participants) | 17 | 18
  Heart rate on Day 3 at 24 hours | 90.8 (15.46) | 95.1 (13.25)
  Heart rate at follow-up Day 7: number analyzed (Participants) | 16 | 15
  Heart rate at follow-up Day 7 | 91.6 (19.06) | 94.2 (15.17)

2. Primary Outcome: Diastolic and Systolic Blood Pressure Assessments Upto Day 7 (Part B)
Description: Vital sign included systolic blood pressure and diastolic blood pressure. Assessments were performed at Pre-dose, 0.5 hours, 2 hours, 6 hours and 12 hours on Day 1, 0 hours on Day 2 at 0 hours, 0.5 hours, 2 hours, 6 hours, 12 hours, 18 hours and 24 hours on Day 3 and at follow-up on Day 7.
Time Frame: Up to Day 7
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of merucry
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
Millimeters of merucry
  Diastolic blood pressure on Day 1 at Pre-dose | 64.7 (12.86) | 53.9 (10.36)
  Diastolic blood pressure on Day 1 at 0.5 hours: number analyzed (Participants) | 20 | 18
  Diastolic blood pressure on Day 1 at 0.5 hours | 64.4 (13.75) | 54.3 (11.39)
  Diastolic blood pressure on Day 1 at 2 hours | 64.4 (12.59) | 54.8 (9.60)
  Diastolic blood pressure on Day 1 at 6 hours | 63.4 (12.08) | 57.1 (9.21)
  Diastolic blood pressure on Day 1 at 12 hours | 64.3 (12.78) | 57.6 (10.05)
  Diastolic blood pressure on Day 2 at 0 hours | 67.0 (15.17) | 57.0 (10.22)
  Diastolic blood pressure on Day 3 at 0 hours: number analyzed (Participants) | 18 | 18
  Diastolic blood pressure on Day 3 at 0 hours | 63.9 (14.50) | 62.7 (14.03)
  Diastolic blood pressure on Day 3 at 0.5 hours: number analyzed (Participants) | 17 | 19
  Diastolic blood pressure on Day 3 at 0.5 hours | 65.6 (13.21) | 61.1 (12.83)
  Diastolic blood pressure on Day 3 at 2 hours: number analyzed (Participants) | 18 | 19
  Diastolic blood pressure on Day 3 at 2 hours | 65.2 (10.34) | 58.1 (11.20)
  Diastolic blood pressure on Day 3 at 6 hours: number analyzed (Participants) | 17 | 19
  Diastolic blood pressure on Day 3 at 6 hours | 65.2 (13.83) | 62.2 (16.59)
  Diastolic blood pressure on Day 3 at 12 hours: number analyzed (Participants) | 18 | 19
  Diastolic blood pressure on Day 3 at 12 hours | 70.0 (16.40) | 60.6 (13.20)
  Diastolic blood pressure on Day 3 at 18 hours: number analyzed (Participants) | 17 | 17
  Diastolic blood pressure on Day 3 at 18 hours | 73.2 (16.31) | 61.8 (10.50)
  Diastolic blood pressure on Day 3 at 24 hours: number analyzed (Participants) | 17 | 18
  Diastolic blood pressure on Day 3 at 24 hours | 66.4 (15.19) | 61.1 (13.06)
  Diastolic blood pressure on follow-up Day 7: number analyzed (Participants) | 16 | 15
  Diastolic blood pressure on follow-up Day 7 | 66.4 (11.58) | 62.7 (8.52)
  Systolic blood pressure on Day 1 at Pre-dose | 122.0 (18.97) | 106.1 (12.68)
  Systolic blood pressure on Day 1 at 0.5 hours: number analyzed (Participants) | 20 | 18
  Systolic blood pressure on Day 1 at 0.5 hours | 118.8 (20.01) | 105.7 (12.66)
  Systolic blood pressure on Day 1 at 2 hours | 122.9 (14.85) | 107.5 (20.49)
  Systolic blood pressure on Day 1 at 6 hours | 121.6 (17.80) | 118.7 (16.41)
  Systolic blood pressure on Day 1 at 12 hours | 122.9 (21.88) | 116.9 (24.33)
  Systolic blood pressure on Day 2 at 0 hours | 131.6 (23.68) | 114.8 (18.94)
  Systolic blood pressure on Day 3 at 0 hours: number analyzed (Participants) | 18 | 18
  Systolic blood pressure on Day 3 at 0 hours | 124.4 (16.32) | 125.2 (23.70)
  Systolic blood pressure on Day 3 at 0.5 hours: number analyzed (Participants) | 17 | 19
  Systolic blood pressure on Day 3 at 0.5 hours | 127.1 (15.76) | 121.9 (23.60)
  Systolic blood pressure on Day 3 at 2 hours: number analyzed (Participants) | 18 | 19
  Systolic blood pressure on Day 3 at 2 hours | 125.2 (14.77) | 118.5 (20.87)
  Systolic blood pressure on Day 3 at 6 hours: number analyzed (Participants) | 17 | 19
  Systolic blood pressure on Day 3 at 6 hours | 127.8 (19.01) | 118.5 (19.60)
  Systolic blood pressure on Day 3 at 12 hours: number analyzed (Participants) | 18 | 19
  Systolic blood pressure on Day 3 at 12 hours | 130.2 (21.95) | 123.2 (24.61)
  Systolic blood pressure on Day 3 at 18 hours: number analyzed (Participants) | 17 | 17
  Systolic blood pressure on Day 3 at 18 hours | 137.5 (23.92) | 129.0 (17.45)
  Systolic blood pressure on Day 3 at 24 hours: number analyzed (Participants) | 17 | 18
  Systolic blood pressure on Day 3 at 24 hours | 128.8 (20.43) | 130.3 (24.97)
  Systolic blood pressure on follow-up Day 7: number analyzed (Participants) | 16 | 15
  Systolic blood pressure on follow-up Day 7 | 129.1 (22.22) | 129.9 (17.92)

3. Primary Outcome: Electrocardiogram (ECG) Parameters, Including PR, QRS, QT, and QTCU and RR Intervals Upto Day 7 (Part B)
Description: Single 12-lead ECGs were obtained using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, and QTCU and RR intervals. Assessments were performed at Pre-dose on Day 1, at 12 hours on Day 3 and at follow-up Day 7.
Time Frame: Up to Day 7
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
millisecond
  PR interval on Day 1,Pre-dose: number analyzed (Participants) | 5 | 8
  PR interval on Day 1,Pre-dose | 136.8 (24.19) | 139.0 (25.09)
  PR interval on Day 3,12 hours: number analyzed (Participants) | 13 | 16
  PR interval on Day 3,12 hours | 128.5 (42.09) | 149.3 (19.76)
  PR interval at follow-up: number analyzed (Participants) | 4 | 13
  PR interval at follow-up | 140.4 (17.81) | 144.8 (20.73)
  QRS duration on Day 1,Pre-dose: number analyzed (Participants) | 5 | 8
  QRS duration on Day 1,Pre-dose | 98.0 (9.27) | 95.5 (16.62)
  QRS duration on Day 3,12 hours: number analyzed (Participants) | 13 | 16
  QRS duration on Day 3,12 hours | 82.8 (8.66) | 98.8 (15.86)
  QRS duration at follow-up Day 7: number analyzed (Participants) | 15 | 13
  QRS duration at follow-up Day 7 | 84.4 (9.01) | 88.6 (16.86)
  Uncorrected QT interval on Day 1,Pre-dose: number analyzed (Participants) | 5 | 8
  Uncorrected QT interval on Day 1,Pre-dose | 350.0 (27.96) | 357.5 (44.13)
  Uncorrected QT interval on Day 3,12 hours: number analyzed (Participants) | 13 | 16
  Uncorrected QT interval on Day 3,12 hours | 357.8 (48.90) | 369.8 (33.92)
  Uncorrected QT interval at follow-up Day 7: number analyzed (Participants) | 15 | 13
  Uncorrected QT interval at follow-up Day 7 | 354.3 (37.12) | 377.5 (49.46)
  Corrected QT interval(Basett) on Day 1,Pre-dose: number analyzed (Participants) | 1 | 4
  Corrected QT interval(Basett) on Day 1,Pre-dose | 463.0 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 469.4 (66.08)
  Corrected QT interval(Basett) on Day 3,12 hours: number analyzed (Participants) | 6 | 6
  Corrected QT interval(Basett) on Day 3,12 hours | 438.9 (13.02) | 468.9 (41.59)
  Corrected QT interval(Basett) at follow-up Day 7: number analyzed (Participants) | 7 | 6
  Corrected QT interval(Basett) at follow-up Day 7 | 453.5 (31.57) | 483.5 (46.51)
  Corrected QT interval(Fridericia), Day 1,Pre-dose: number analyzed (Participants) | 1 | 4
  Corrected QT interval(Fridericia), Day 1,Pre-dose | 423.4 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 418.1 (49.03)
  Corrected QT interval(Fridericia), Day 3,12 hours: number analyzed (Participants) | 6 | 6
  Corrected QT interval(Fridericia), Day 3,12 hours | 406.3 (20.18) | 432.7 (35.92)
  Corrected QT interval(Fridericia),follow-up Day 7: number analyzed (Participants) | 7 | 6
  Corrected QT interval(Fridericia),follow-up Day 7 | 419.5 (12.66) | 439.6 (36.29)
  QTCU on Day 1,Pre-dose: number analyzed (Participants) | 4 | 4
  QTCU on Day 1,Pre-dose | 458.3 (8.81) | 447.3 (27.65)
  QTCU on Day 3,12 hours: number analyzed (Participants) | 7 | 10
  QTCU on Day 3,12 hours | 440.3 (40.07) | 445.4 (28.11)
  QTCU at follow-up Day 7: number analyzed (Participants) | 8 | 7
  QTCU at follow-up Day 7 | 441.6 (17.72) | 457.3 (26.12)
  RR interval on Day 1,Pre-dose: number analyzed (Participants) | 1 | 4
  RR interval on Day 1,Pre-dose | 584.6 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 513.6 (97.25)
  RR interval on Day 3,12 hours: number analyzed (Participants) | 6 | 6
  RR interval on Day 3,12 hours | 638.8 (135.85) | 623.2 (76.02)
  RR interval at follow-up Day 7: number analyzed (Participants) | 7 | 6
  RR interval at follow-up Day 7 | 661.7 (203.97) | 582.9 (128.96)

4. Primary Outcome: Hematology Parameters Basophils, Eosinophil, Lymphocytes, Monocytes, Total Neutrophils, Platelet Count and White Blood Cell Count Upto Day 7 (Part B)
Description: Hematology parameters included basophils, eosinophil, lymphocytes, monocytes, total neutrophils, platelet count and white blood cell count. Assessments were performed at Pre-dose on Day 1, at 12 hours on Day 3 and at follow-up Day 7.
Time Frame: Up to Day 7
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: giga per liter
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
giga per liter
  Basophils on Day 1 at Pre-dose: number analyzed (Participants) | 1 | 3
  Basophils on Day 1 at Pre-dose | 0.020 (NA) — Standard deviation was not calculated as a single participant was analyzed. | 0.000 (0.0000)
  Basophils on Day 3 at 12 hours: number analyzed (Participants) | 13 | 15
  Basophils on Day 3 at 12 hours | 0.015 (0.0296) | 0.011 (0.0277)
  Basophils on Follow-up Day 7: number analyzed (Participants) | 9 | 11
  Basophils on Follow-up Day 7 | 0.025 (0.0431) | 0.113 (0.1848)
  Eosinophils on Day 1 at Pre-dose: number analyzed (Participants) | 1 | 3
  Eosinophils on Day 1 at Pre-dose | 0.110 (NA) — Standard deviation was not calculated as a single participant was analyzed. | 0.233 (0.4041)
  Eosinophils on Day 3 at 12 hours: number analyzed (Participants) | 13 | 15
  Eosinophils on Day 3 at 12 hours | 0.096 (0.1624) | 0.163 (0.2280)
  Eosinophils on Follow-up Day 7: number analyzed (Participants) | 9 | 11
  Eosinophils on Follow-up Day 7 | 0.137 (0.1074) | 0.324 (0.4957)
  Lymphocytes on Day 1 at Pre-dose: number analyzed (Participants) | 2 | 3
  Lymphocytes on Day 1 at Pre-dose | 4.81 (4.603) | 0.52 (0.266)
  Lymphocytes on Day 3 at 12 hours: number analyzed (Participants) | 14 | 15
  Lymphocytes on Day 3 at 12 hours | 1.08 (0.948) | 0.60 (0.380)
  Lymphocytes on Follow-up Day 7: number analyzed (Participants) | 12 | 11
  Lymphocytes on Follow-up Day 7 | 1.61 (1.244) | 1.04 (0.663)
  Monocytes on Day 1 at Pre-dose: number analyzed (Participants) | 2 | 3
  Monocytes on Day 1 at Pre-dose | 1.760 (1.7112) | 0.377 (0.3356)
  Monocytes on Day 3 at 12 hours: number analyzed (Participants) | 14 | 15
  Monocytes on Day 3 at 12 hours | 0.503 (0.4046) | 0.571 (0.6336)
  Monocytes on Follow-up Day 7: number analyzed (Participants) | 11 | 11
  Monocytes on Follow-up Day 7 | 0.669 (0.3986) | 0.727 (0.5812)
  Total neutrophils on Day 1 at Pre-dose: number analyzed (Participants) | 2 | 3
  Total neutrophils on Day 1 at Pre-dose | 6.990 (4.5113) | 7.807 (9.3471)
  Total neutrophils on Day 3 at 12 hours: number analyzed (Participants) | 4 | 15
  Total neutrophils on Day 3 at 12 hours | 11.563 (6.0785) | 9.931 (6.8583)
  Total neutrophils on Follow-up Day 7: number analyzed (Participants) | 11 | 11
  Total neutrophils on Follow-up Day 7 | 16.775 (21.6419) | 11.761 (5.5496)
  Platelet count on Day 1 at Pre-dose: number analyzed (Participants) | 6 | 4
  Platelet count on Day 1 at Pre-dose | 170.3 (67.26) | 236.0 (158.73)
  Platelet count on Day 3 at 12 hours: number analyzed (Participants) | 18 | 18
  Platelet count on Day 3 at 12 hours | 218.9 (120.68) | 235.9 (134.43)
  Platelet count on Follow-up Day 7: number analyzed (Participants) | 16 | 14
  Platelet count on Follow-up Day 7 | 334.1 (169.06) | 369.8 (169.70)
  White blood cell count on Day 1 at Pre-dose: number analyzed (Participants) | 6 | 4
  White blood cell count on Day 1 at Pre-dose | 15.15 (14.289) | 10.72 (8.829)
  White blood cell count on Day 3 at 12 hours: number analyzed (Participants) | 18 | 18
  White blood cell count on Day 3 at 12 hours | 14.82 (5.927) | 11.82 (6.618)
  White blood cell count on Follow-up Day 7: number analyzed (Participants) | 16 | 14
  White blood cell count on Follow-up Day 7 | 14.09 (5.197) | 36.56 (84.293)

5. Primary Outcome: Hematology Parameters Red Blood Cell Count and Reticulocyte Count Assessment Upto Day 7 (Part B)
Description: Hematology parameters included red blood cell count and reticulocyte count. Assessments were performed at Pre-dose on Day 1, at 12 hours on Day 3 and at follow-up Day 7.
Time Frame: Up to Day 7
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: trillion cells per liter
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
trillion cells per liter
  Red blood cell count on Day 1 at Pre-dose: number analyzed (Participants) | 6 | 4
  Red blood cell count on Day 1 at Pre-dose | 3.207 (0.7733) | 2.678 (0.5117)
  Red blood cell count on Day 3 at 12 hours: number analyzed (Participants) | 18 | 18
  Red blood cell count on Day 3 at 12 hours | 3.271 (0.5725) | 3.076 (0.5001)
  Red blood cell count on Follow-up Day 7: number analyzed (Participants) | 16 | 14
  Red blood cell count on Follow-up Day 7 | 3.352 (0.6374) | 3.314 (0.7700)
  Reticulocyte count on Day 1 at Pre-dose: number analyzed (Participants) | 3 | 1
  Reticulocyte count on Day 1 at Pre-dose | 0.025 (0.0195) | 0.044 (NA) — Standard deviation was not calculated as a single participant was analyzed.
  Reticulocyte count on Day 3 at 12 hours: number analyzed (Participants) | 10 | 12
  Reticulocyte count on Day 3 at 12 hours | 0.832 (2.5186) | 3.697 (12.6920)
  Reticulocyte count on Follow-up Day 7: number analyzed (Participants) | 11 | 9
  Reticulocyte count on Follow-up Day 7 | 1.607 (5.1055) | 8.629 (25.6392)

6. Primary Outcome: Hematology Parameter Hemoglobin and Mean Corpuscle Hemoglobin Concentration (MCHC) Assessment Upto Day 7 (Part B)
Description: Hematology parameters included hemoglobin and MCHC. Assessments were performed at Pre-dose on Day 1, at 12 hours on Day 3 and at follow-up Day 7.
Time Frame: Up to Day 7
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
grams per liter
  Hemoglobin on Day 1 at Pre-dose: number analyzed (Participants) | 6 | 4
  Hemoglobin on Day 1 at Pre-dose | 99.5 (24.83) | 84.0 (13.09)
  Hemoglobin on Day 3 at 12 hours: number analyzed (Participants) | 18 | 18
  Hemoglobin on Day 3 at 12 hours | 195.8 (286.77) | 180.8 (266.16)
  Hemoglobin on Follow-up Day 7: number analyzed (Participants) | 16 | 14
  Hemoglobin on Follow-up Day 7 | 244.7 (401.03) | 213.6 (301.50)
  MCHC on Day 1 at Pre-dose: number analyzed (Participants) | 6 | 4
  MCHC on Day 1 at Pre-dose | 331.8 (10.68) | 339.5 (19.12)
  MCHC on Day 3 at 12 hours: number analyzed (Participants) | 17 | 16
  MCHC on Day 3 at 12 hours | 328.4 (14.73) | 330.8 (16.82)
  MCHC on Follow-up Day 7: number analyzed (Participants) | 15 | 11
  MCHC on Follow-up Day 7 | 327.8 (12.35) | 325.4 (6.82)

7. Primary Outcome: Hematology Parameter Mean Corpuscle Volume (MCV) Assessment Upto Day 7 (Part B)
Description: Hematology parameter included MCV. Assessments were performed at Pre-dose on Day 1, at 12 hours on Day 3 and at follow-up Day 7.
Time Frame: Up to Day 7
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
femtoliters
  MCV on Day 1 at Pre-dose: number analyzed (Participants) | 6 | 3
  MCV on Day 1 at Pre-dose | 77.37 (33.654) | 93.87 (0.971)
  MCV on Day 3 at 12 hours: number analyzed (Participants) | 18 | 17
  MCV on Day 3 at 12 hours | 91.28 (5.611) | 90.69 (5.976)
  MCV on Follow-up Day 7: number analyzed (Participants) | 16 | 13
  MCV on Follow-up Day 7 | 92.53 (7.234) | 90.46 (7.063)

8. Primary Outcome: Hematology Parameter Mean Corpuscle Hemoglobin (MCH) Assessment Upto Day 7 (Part B)
Description: Hematology parameter included MCH. Assessments were performed at Pre-dose on Day 1, at 12 hours on Day 3 and at follow-up Day 7.
Time Frame: Up to Day 7
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: picograms
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
picograms
  MCH on Day 1 at Pre-dose: number analyzed (Participants) | 3 | 3
  MCH on Day 1 at Pre-dose | 30.30 (4.493) | 30.40 (0.361)
  MCH on Day 3 at 12 hours: number analyzed (Participants) | 13 | 11
  MCH on Day 3 at 12 hours | 30.02 (2.695) | 30.32 (1.955)
  MCH on Follow-up Day 7: number analyzed (Participants) | 11 | 8
  MCH on Follow-up Day 7 | 30.49 (2.545) | 30.25 (2.071)

9. Primary Outcome: Hematology Parameter Hematocrit Assessment Upto Day 7 (Part B)
Description: Hematology parameter included hematocrit. Assessments were performed at Pre-dose on Day 1, at 12 hours on Day 3 and at follow-up Day 7.
Time Frame: Up to Day 7
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Fraction
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
Fraction
  Hematocrit on Day 1 at Pre-dose: number analyzed (Participants) | 6 | 4
  Hematocrit on Day 1 at Pre-dose | 0.201 (0.1666) | 0.196 (0.1333)
  Hematocrit on Day 3 at 12 hours: number analyzed (Participants) | 18 | 18
  Hematocrit on Day 3 at 12 hours | 0.271 (0.1071) | 1.519 (5.3867)
  Hematocrit on Follow-up Day 7: number analyzed (Participants) | 16 | 14
  Hematocrit on Follow-up Day 7 | 0.254 (0.1298) | 2.270 (7.5504)

10. Primary Outcome: Clinical Chemistry Parameters Calcium, Chloride, Carbon Dioxide, Glucose, Potassium, Sodium, Urea/Blood Urea Nitrogen Assessment Upto Day 7 (Part B)
Description: Clinical chemistry parameters included calcium, chloride, carbon dioxide, glucose, potassium, sodium, Urea/Blood urea nitrogen. Assessments were performed at Pre-dose on Day 1, at 12 hours on Day 3 and at follow-up Day 7.
Time Frame: Up to Day 7
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: millimoles per liter
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
millimoles per liter
  Calcium on Day 1 at Pre-dose: number analyzed (Participants) | 3 | 5
  Calcium on Day 1 at Pre-dose | 1.927 (0.0736) | 1.894 (0.1070)
  Calcium on Day 3 at 12 hours: number analyzed (Participants) | 11 | 13
  Calcium on Day 3 at 12 hours | 1.983 (0.1220) | 1.982 (0.1296)
  Calcium on Follow-up Day 7: number analyzed (Participants) | 12 | 11
  Calcium on Follow-up Day 7 | 2.155 (0.1016) | 2.104 (0.1448)
  Chloride on Day 1 at Pre-dose: number analyzed (Participants) | 5 | 5
  Chloride on Day 1 at Pre-dose | 108.8 (5.93) | 104.0 (7.18)
  Chloride on Day 3 at 12 hours: number analyzed (Participants) | 18 | 18
  Chloride on Day 3 at 12 hours | 107.7 (5.12) | 106.0 (6.05)
  Chloride on Follow-up Day 7: number analyzed (Participants) | 16 | 15
  Chloride on Follow-up Day 7 | 104.4 (3.76) | 103.7 (5.01)
  Carbon dioxide on Day 1 at Pre-dose: number analyzed (Participants) | 5 | 5
  Carbon dioxide on Day 1 at Pre-dose | 24.40 (5.273) | 23.28 (6.685)
  Carbon dioxide on Day 3 at 12 hours: number analyzed (Participants) | 18 | 18
  Carbon dioxide on Day 3 at 12 hours | 26.35 (3.176) | 27.83 (6.071)
  Carbon dioxide on Follow-up Day 7: number analyzed (Participants) | 16 | 15
  Carbon dioxide on Follow-up Day 7 | 27.69 (3.728) | 27.39 (3.412)
  Glucose on Day 1 at Pre-dose: number analyzed (Participants) | 5 | 5
  Glucose on Day 1 at Pre-dose | 6.015 (0.7499) | 6.159 (1.1230)
  Glucose on Day 3 at 12 hours: number analyzed (Participants) | 18 | 18
  Glucose on Day 3 at 12 hours | 8.095 (2.1569) | 7.411 (1.6158)
  Glucose on Follow-up Day 7: number analyzed (Participants) | 15 | 15
  Glucose on Follow-up Day 7 | 6.701 (1.6354) | 7.285 (1.5159)
  Potassium on Day 1 at Pre-dose: number analyzed (Participants) | 5 | 5
  Potassium on Day 1 at Pre-dose | 3.88 (0.444) | 3.72 (0.164)
  Potassium on Day 3 at 12 hours: number analyzed (Participants) | 18 | 18
  Potassium on Day 3 at 12 hours | 4.20 (0.511) | 3.96 (0.578)
  Potassium on Follow-up Day 7: number analyzed (Participants) | 16 | 15
  Potassium on Follow-up Day 7 | 3.83 (0.505) | 3.92 (0.435)
  Sodium on Day 1 at Pre-dose: number analyzed (Participants) | 5 | 5
  Sodium on Day 1 at Pre-dose | 141.8 (3.11) | 137.6 (3.71)
  Sodium on Day 3 at 12 hours: number analyzed (Participants) | 18 | 18
  Sodium on Day 3 at 12 hours | 143.1 (4.46) | 141.6 (4.03)
  Sodium on Follow-up Day 7: number analyzed (Participants) | 16 | 15
  Sodium on Follow-up Day 7 | 141.9 (4.59) | 139.7 (4.58)
  Urea/Blood urea nitrogen on Day 1 at Pre-dose: number analyzed (Participants) | 5 | 5
  Urea/Blood urea nitrogen on Day 1 at Pre-dose | 6.433 (3.0512) | 11.399 (7.4163)
  Urea/Blood urea nitrogen on Day 3 at 12 hours: number analyzed (Participants) | 18 | 18
  Urea/Blood urea nitrogen on Day 3 at 12 hours | 10.410 (6.5542) | 9.485 (6.5777)
  Urea/Blood urea nitrogen on Follow-up Day 7: number analyzed (Participants) | 16 | 15
  Urea/Blood urea nitrogen on Follow-up Day 7 | 11.787 (9.3546) | 9.207 (6.5375)

11. Primary Outcome: Clinical Chemistry Parameters Direct Bilirubin, Total Bilirubin, Creatinine and Uric Acid Assessment Upto Day 7 (Part B)
Description: Clinical chemistry parameters included direct bilirubin, total bilirubin, creatinine and uric acid. Assessments were performed at Pre-dose on Day 1, at 12 hours on Day 3 and at follow-up Day 7.
Time Frame: Up to Day 7
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
micromoles per liter
  Direct bilirubin on Day 1 at Pre-dose: number analyzed (Participants) | 4 | 5
  Direct bilirubin on Day 1 at Pre-dose | 10.663 (7.8146) | 13.792 (17.7932)
  Direct bilirubin on Day 3 at 12 hours: number analyzed (Participants) | 15 | 16
  Direct bilirubin on Day 3 at 12 hours | 10.446 (14.2406) | 10.428 (22.4573)
  Direct bilirubin on Follow-up Day 7: number analyzed (Participants) | 12 | 11
  Direct bilirubin on Follow-up Day 7 | 4.140 (3.5564) | 2.576 (1.6103)
  Total bilirubin on Day 1 at Pre-dose: number analyzed (Participants) | 5 | 5
  Total bilirubin on Day 1 at Pre-dose | 16.672 (11.1375) | 21.926 (20.4768)
  Total bilirubin on Day 3 at 12 hours: number analyzed (Participants) | 17 | 17
  Total bilirubin on Day 3 at 12 hours | 16.803 (15.8462) | 14.119 (24.8465)
  Total bilirubin on Follow-up Day 7: number analyzed (Participants) | 14 | 12
  Total bilirubin on Follow-up Day 7 | 12.547 (10.7837) | 5.818 (3.0149)
  Creatinine on Day 1 at Pre-dose: number analyzed (Participants) | 5 | 5
  Creatinine on Day 1 at Pre-dose | 85.194 (19.9261) | 126.228 (71.9085)
  Creatinine on Day 3 at 12 hours: number analyzed (Participants) | 18 | 18
  Creatinine on Day 3 at 12 hours | 108.189 (102.4388) | 103.066 (90.6252)
  Creatinine on Follow-up Day 7: number analyzed (Participants) | 16 | 15
  Creatinine on Follow-up Day 7 | 91.726 (45.2713) | 90.516 (71.8052)
  Uric acid on Day 1 at Pre-dose: number analyzed (Participants) | 3 | 3
  Uric acid on Day 1 at Pre-dose | 233.432 (67.9909) | 181.453 (203.5924)
  Uric acid on Day 3 at 12 hours: number analyzed (Participants) | 13 | 13
  Uric acid on Day 3 at 12 hours | 192.925 (143.7971) | 228.144 (134.9558)
  Uric acid on Follow-up Day 7: number analyzed (Participants) | 12 | 12
  Uric acid on Follow-up Day 7 | 241.766 (72.0137) | 225.326 (144.4626)

12. Primary Outcome: Clinical Chemistry Parameters Alkaline Phosphatase, Asparatate Amino Transferase, Alanine Amino Transferase, Gamma Glutamyl Transferase Assessment Upto Day 7 (Part B)
Description: Clinical chemistry parameters included alkaline phosphatase, asparatate amino transferase, alanine amino transferase, gamma glutamyl transferase. Assessments were performed at Pre-dose on Day 1, at 12 hours on Day 3 and at follow-up Day 7.
Time Frame: Up to Day 7
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
International units per liter
  Alkaline phosphatase on Day 1 at Pre-dose: number analyzed (Participants) | 5 | 5
  Alkaline phosphatase on Day 1 at Pre-dose | 76.6 (18.57) | 94.0 (50.86)
  Alkaline phosphatase on Day 3 at 12 hours: number analyzed (Participants) | 17 | 17
  Alkaline phosphatase on Day 3 at 12 hours | 130.9 (68.16) | 109.2 (63.02)
  Alkaline phosphatase on Follow-up Day 7: number analyzed (Participants) | 14 | 12
  Alkaline phosphatase on Follow-up Day 7 | 101.1 (40.15) | 117.0 (56.07)
  Alanine amino transferase on Day 1 at Pre-dose: number analyzed (Participants) | 5 | 5
  Alanine amino transferase on Day 1 at Pre-dose | 101.8 (105.98) | 56.8 (42.20)
  Alanine amino transferase on Day 3 at 12 hours: number analyzed (Participants) | 17 | 17
  Alanine amino transferase on Day 3 at 12 hours | 73.4 (71.27) | 43.6 (50.72)
  Alanine amino transferase on Follow-up Day 7: number analyzed (Participants) | 14 | 12
  Alanine amino transferase on Follow-up Day 7 | 44.9 (42.74) | 117.9 (224.94)
  Asparatate amino transferase on Day 1 at Pre-dose: number analyzed (Participants) | 5 | 5
  Asparatate amino transferase on Day 1 at Pre-dose | 96.8 (46.09) | 64.6 (37.14)
  Asparatate amino transferase on Day 3 at 12 hours: number analyzed (Participants) | 17 | 17
  Asparatate amino transferase on Day 3 at 12 hours | 56.2 (34.60) | 62.0 (71.54)
  Asparatate amino transferase on Follow-up Day 7: number analyzed (Participants) | 14 | 12
  Asparatate amino transferase on Follow-up Day 7 | 35.6 (20.25) | 76.5 (106.39)
  Gamma glutamyl transferase on Day 1 at Pre-dose: number analyzed (Participants) | 2 | 3
  Gamma glutamyl transferase on Day 1 at Pre-dose | 96.0 (22.63) | 40.7 (25.89)
  Gamma glutamyl transferase on Day 3 at 12 hours: number analyzed (Participants) | 13 | 12
  Gamma glutamyl transferase on Day 3 at 12 hours | 156.5 (149.89) | 98.4 (71.85)
  Gamma glutamyl transferase on Follow-up Day 7: number analyzed (Participants) | 11 | 12
  Gamma glutamyl transferase on Follow-up Day 7 | 116.4 (105.36) | 143.0 (138.22)

13. Primary Outcome: Clinical Chemistry Parameters Albumin and Total Protein Assessment Upto Day 7 (Part B)
Description: Clinical chemistry parameters included albumin and total protein. Assessments were performed at Pre-dose on Day 1, at 12 hours on Day 3 and at follow-up Day 7.
Time Frame: Up to Day 7
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
grams per liter
  Albumin on Day 1 at Pre-dose: number analyzed (Participants) | 5 | 5
  Albumin on Day 1 at Pre-dose | 25.6 (2.19) | 18.6 (3.21)
  Albumin on Day 3 at 12 hours: number analyzed (Participants) | 17 | 17
  Albumin on Day 3 at 12 hours | 25.5 (5.05) | 22.3 (4.88)
  Albumin on Follow-up Day 7: number analyzed (Participants) | 14 | 12
  Albumin on Follow-up Day 7 | 27.9 (6.62) | 25.5 (6.27)
  Total protein on Day 1 at Pre-dose: number analyzed (Participants) | 5 | 5
  Total protein on Day 1 at Pre-dose | 54.60 (5.983) | 50.20 (2.775)
  Total protein on Day 3 at 12 hours: number analyzed (Participants) | 16 | 17
  Total protein on Day 3 at 12 hours | 55.06 (7.122) | 52.12 (7.457)
  Total protein on Follow-up Day 7: number analyzed (Participants) | 14 | 11
  Total protein on Follow-up Day 7 | 60.86 (8.646) | 58.18 (10.323)

14. Primary Outcome: Number of Participant With Adverse Event (AE) and Serious Adverse Event (SAE) Assessment Upto Day 7 (Part A)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed in the definition above, or is an event of possible drug-induced liver injury.
Time Frame: Up to Day 7
Population: The All Subjects - Part A Population was defined as all participants in Part A who received at least one dose of study medication.
Measure: Number; unit: Participants
Groups:
- Part A: Eligible participants received multiple single intravenous escalating doses of GSK2586881 (0.1 milligrams per kg [mg/kg], 0.2 mg/kg, 0.4 mg/kg, 0.8 mg/kg) as a slow infusion over 3-5 minutes over 2 days.
Arm/Group | Part A
Number analyzed (Participants) | 5
Participants
  Any AE | 5
  Anys SAE | 3

15. Primary Outcome: Number of Par With AE and Serious Adverse Event (SAE) Assessment Upto Day 7 (Part B)
Description: as for outcome 14
Time Frame: Up to Day 7
Population: All Subjects - Part B Population.
Measure: Number; unit: Participant
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
Participant
  Any AE | 14 | 15
  Any SAE | 4 | 3

16. Secondary Outcome: Analysis of GSK2586881 Plasma Pharmacokinetic Concentration (Part A)
Description: Blood samples for pharmacokinetic analysis of GSK2586881 were collected Pre-dose, 5 minutes, 10 minutes, 2 hours, 6 hours, 10 hours, 12 hours (Day 1), 0 hours, 1 hour, 12 hours, 24 hours (Day 2). Data has been presented for GSK2586881 Plasma Pharmacokinetic Concentration versus time data for Part A
Time Frame: Pre-dose, 5 minutes, 10 minutes, 2 hours, 6 hours, 10 hours, 12 hours (Day 1), 0 hours, 1 hour, 12 hours, 24 hours (Day 2)
Population: The Pharmacokinetic - Part A Population was defined as participants in the All Subjects - Part A population for whom a pharmacokinetic sample was obtained and analyzed and a result reported and received an active dose of GSK2586881.
Measure: Mean (Standard Deviation); unit: nano grams per milliliter
Arm/Group | Part A
Number analyzed (Participants) | 5
nano grams per milliliter
  GSK2586881 concentration at Pre-dose on Day 1 | NA (NA) — No concentration values detected for Pre-dose.
  GSK2586881 concentration at 5 minutes on Day 1 | 2854.0 (595.47)
  GSK2586881 concentration at 10 minutes on Day 1 | 2692.8 (629.78)
  GSK2586881 concentration at 2 hours on Day 1 | 2047.4 (497.19)
  GSK2586881 concentration at 6 hours on Day 1 | 5460.0 (3213.96)
  GSK2586881 concentration at 10 hours on Day 1 | 10276.6 (2641.49)
  GSK2586881 concentration at 12 hours on Day 1 | 8265.4 (1905.29)
  GSK2586881 concentration at 0 hours on Day 2 | 3621.6 (2654.21)
  GSK2586881 concentration at 1 hour on Day 2 | 17558.6 (4359.04)
  GSK2586881 concentration at 12 hours on Day 2 | 7237.8 (4281.27)
  GSK2586881 concentration at 24 hours on Day 2 | 3517.8 (2433.49)

17. Secondary Outcome: Analysis of GSK2586881 Plasma Pharmacokinetic Concentration (Part B)
Description: Blood samples for pharmacokinetic analysis of GSK2586881 were collected Pre-dose, 0.5 Hours, 2 hours, 6 hours, 12 hours (Day 1), 0 hours (Day 2), 0 hours, 0.5 hours, 2 hours, 6 hours, 12 hours, 18 hours and 24 hours (Day 3). Data has been presented for GSK2586881 Plasma Pharmacokinetic Concentration versus time data for Part B.
Time Frame: Pre-dose, 0.5 Hours, 2 hours, 6 hours, 12 hours (Day 1), 0 hours (Day 2), 0 hours, 0.5 hours, 2 hours, 6 hours, 12 hours, 18 hours and 24 hours (Day 3)
Population: The Pharmacokinetic - Part B Population was defined as participants in the All Subjects - Part B population for whom a pharmacokinetic sample was obtained and analyzed and a result reported and received an active dose of GSK2586881. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Part B (GSK2586881 BID)
Number analyzed (Participants) | 19
nanograms per milliliter
  GSK2586881 concentration at Pre-dose on Day 1 | NA (NA) — No concentration values detected for Pre-dose.
  GSK2586881 concentration at 0.5 hours on Day 1 | 5489.3 (1727.81)
  GSK2586881 concentration at 2 hours on Day 1: number analyzed (Participants) | 18
  GSK2586881 concentration at 2 hours on Day 1 | 4334.0 (1880.42)
  GSK2586881 concentration at 6 hours on Day 1 | 5065.4 (8679.92)
  GSK2586881 concentration at 12 hours on Day 1: number analyzed (Participants) | 17
  GSK2586881 concentration at 12 hours on Day 1 | 1815.9 (809.52)
  GSK2586881 concentration at 0 hours on Day 2: number analyzed (Participants) | 18
  GSK2586881 concentration at 0 hours on Day 2 | 2115.3 (1164.12)
  GSK2586881 concentration at 0 hours on Day 3: number analyzed (Participants) | 18
  GSK2586881 concentration at 0 hours on Day 3 | 2306.6 (1356.75)
  GSK2586881 concentration at 0.5 hours on Day 3: number analyzed (Participants) | 18
  GSK2586881 concentration at 0.5 hours on Day 3 | 6810.4 (3135.66)
  GSK2586881 concentration at 2 hours on Day 3 | 6060.7 (2956.33)
  GSK2586881 concentration at 6 hours on Day 3: number analyzed (Participants) | 17
  GSK2586881 concentration at 6 hours on Day 3 | 3808.9 (1953.82)
  GSK2586881 concentration at 12 hours on Day 3: number analyzed (Participants) | 18
  GSK2586881 concentration at 12 hours on Day 3 | 2416.6 (1601.08)
  GSK2586881 concentration at 18 hours on Day 3: number analyzed (Participants) | 16
  GSK2586881 concentration at 18 hours on Day 3 | 2701.6 (1874.28)
  GSK2586881 concentration at 24 hours on Day 3: number analyzed (Participants) | 16
  GSK2586881 concentration at 24 hours on Day 3 | 2254.7 (1233.58)

18. Secondary Outcome: Analysis of Pharmacokinetic Parameter Clearance (CL) for GSK2586881 (Part A)
Description: Blood samples for pharmacokinetic analysis of GSK2586881 were collected at Pre-dose, 0 hour, 5 minutes, 10 minutes, 2 hours, 6 hours, 10 hours, 12 hours, 24 hours, 25 hours, 36 hours and 48 hours. CL was defined as the systemic clearance of parent drug. Clearance was calculated for individual participant and geometric mean of the values from all participants was reported.
Time Frame: Pre-dose, 0 hour, 5 minutes, 10 minutes, 2 hours, 6 hours, 10 hours, 12 hours, 24 hours, 25 hours, 36 hours, 48 hours
Population: Pharmacokinetic - Part A Population.
Measure: Geometric Mean (Standard Error); unit: liters per hour
Arm/Group | Part A
Number analyzed (Participants) | 5
liters per hour | 0.384 (0.0886)

19. Secondary Outcome: Analysis Pharmacokinetic Parameter Clearance (CL) for GSK2586881 (Part B)
Description: as for outcome 18
Time Frame: Pre-dose, 0 hour, 5 minutes, 10 minutes, 2 hours, 6 hours, 10 hours, 12 hours, 24 hours, 25 hours, 36 hours, 48 hours
Population: Pharmacokinetic - Part B Population.
Measure: Geometric Mean (Standard Error); unit: liters per hour
Arm/Group | Part B (GSK2586881 BID)
Number analyzed (Participants) | 19
liters per hour | 0.698 (0.0608)

20. Secondary Outcome: Pharmacodynamic/Biomarker Analysis (Renin-angiotensin System Cascade Biomarkers) to Include Angiotensin (Ang) II and Ang (1-7) Upto Day 2 (Part A)
Description: Renin-angiotensin system cascade biomarkers included Ang II and Ang (1-7). Blood samples for biomarker analyses were collected at Pre-dose, 5 minutes, 10 minutes, 2 hours, 6 hours, 10 hours, 12 hours (Day 1) and 0 hours, 1 hour, 12 hours and 24 hours on Day 2.
Time Frame: Pre-dose, 5 minutes, 10 minutes, 2 hours, 6 hours, 10 hours, 12 hours (Day 1) and 0 hours, 1 hour, 12 hours and 24 hours (Day 2).
Population: All Subjects - Part A Population
Measure: Geometric Mean (95% Confidence Interval); unit: picograms per milliliter
Arm/Group | Part A
Number analyzed (Participants) | 5
picograms per milliliter
  AngII at Pre-dose on Day 1 | 26.5 [14.0 to 50.1]
  AngII at 5 minutes on Day 1 | 7.7 [3.2 to 18.4]
  AngII at 10 minutes on Day 1 | 6.2 [3.4 to 11.3]
  AngII at 2 hours on Day 1 | 3.9 [0.9 to 17.4]
  AngII at 6 hours on Day 1 | 4.3 [0.8 to 22.3]
  AngII at 10 hours on Day 1 | 2.0 [0.4 to 10.3]
  AngII at 12 hours on Day 1 | 3.3 [0.8 to 13.9]
  AngII at 0 hours on Day 2 | 1.7 [0.2 to 13.3]
  AngII at 1 hour on Day 2 | 4.3 [0.3 to 70.9]
  AngII at 12 hours on Day 2 | 1.8 [0.2 to 15.5]
  AngII at 24 hours on Day 2 | 1.5 [0.2 to 10.5]
  Ang1-7 at Pre-dose on Day 1 | 4.3 [0.9 to 21.4]
  Ang1-7 at 5 minutes on Day 1 | 28.7 [10.9 to 75.8]
  Ang1-7 at 10 minutes on Day 1 | 25.7 [11.6 to 56.8]
  Ang1-7 at 2 hours on Day 1 | 18.7 [6.4 to 54.1]
  Ang1-7 at 6 hours on Day 1 | 22.8 [5.3 to 97.9]
  Ang1-7 at 10 hours on Day 1 | 16.8 [1.2 to 243.5]
  Ang1-7 at 12 hours on Day 1 | 15.1 [1.2 to 183.2]
  Ang1-7 at 0 hours on Day 2 | 9.1 [0.6 to 130.1]
  Ang1-7 at 1 hour on Day 2 | 20.9 [1.3 to 331.3]
  Ang1-7 at 12 hours on Day 2 | 18.8 [2.6 to 138.4]
  Ang1-7 at 24 hours on Day 2 | 5.2 [0.2 to 122.2]

21. Secondary Outcome: Pharmacodynamic/Biomarker Analysis (Renin-angiotensin System Cascade Biomarkers) to Include Ang II/ Ang (1-7) Upto Day 2 (Part A)
Description: Renin-angiotensin system cascade biomarkers included Ang II/Ang (1-7). Blood samples for biomarker analyses were collected at Pre-dose, 5 minutes, 10 minutes, 2 hours, 6 hours, 10 hours, 12 hours on Day 1 and 0 hours, 1 hour, 12 hours and 24 hours on Day 2.
Time Frame: as for outcome 20
Population: All Subjects - Part A Population.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Part A
Number analyzed (Participants) | 5
Ratio
  AngII/ Ang1-7 at Pre-dose on Day 1 | 6.167 [1.372 to 27.721]
  AngII/ Ang1-7 at 5 minutes on Day 1 | 0.268 [0.099 to 0.722]
  AngII/ Ang1-7 at 10 minutes on Day 1 | 0.241 [0.095 to 0.608]
  AngII/ Ang1-7 at 2 hours on Day 1 | 0.210 [0.036 to 1.226]
  AngII/ Ang1-7 at 6 hours on Day 1 | 0.190 [0.032 to 1.138]
  AngII/ Ang1-7 at 10 hours on Day 1 | 0.118 [0.024 to 0.583]
  AngII/ Ang1-7 at 12 hours on Day 1 | 0.221 [0.012 to 3.959]
  AngII/ Ang1-7 at 0 hours on Day 2 | 0.182 [0.018 to 1.831]
  AngII/ Ang1-7 at 1 hour on Day 2 | 0.206 [0.017 to 2.421]
  AngII/ Ang1-7 at 12 hours on Day 2 | 0.094 [0.007 to 1.268]
  AngII/ Ang1-7 at 24 hours on Day 2 | 0.290 [0.030 to 2.801]

22. Secondary Outcome: Pharmacodynamic/Biomarker Analysis (Renin-angiotensin System Cascade Biomarkers) to Include Ang II, Ang (1-7) and Ang (1-5) Upto Day 5(Part B)
Description: Renin-angiotensin system cascade biomarkers included Ang II, Ang (1-7) and Ang (1-5). Blood samples for biomarker analyses were collected 0.5 hours, 2 hours, 6 hours, 12 hours, 24 hours, 48 hours, 48.5 hours, 50 hours, 54 hours, 60 hours, 66 hours, 72 hours, 96 hours and 120 hours upto Day 5. Data has been presented for median along with the 95% credible interval.
Time Frame: 0.5 hours, 2 hours, 6 hours, 12 hours, 24 hours, 48 hours, 48.5 hours, 50 hours, 54 hours, 60 hours, 66 hours, 72 hours, 96 hours and 120 hours upto Day 5.
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Median (95% Confidence Interval); unit: picograms per milliliter
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
picograms per milliliter
  AngII at 0.5 hours: number analyzed (Participants) | 16 | 18
  AngII at 0.5 hours | 14.14 [7.890 to 25.065] | 2.44 [1.400 to 4.095]
  AngII at 2 hours: number analyzed (Participants) | 16 | 16
  AngII at 2 hours | 12.05 [6.658 to 21.146] | 2.80 [1.585 to 4.735]
  AngII at 6 hours: number analyzed (Participants) | 16 | 15
  AngII at 6 hours | 11.00 [6.084 to 19.518] | 2.89 [1.620 to 4.997]
  AngII at 12 hours: number analyzed (Participants) | 14 | 15
  AngII at 12 hours | 10.90 [5.920 to 19.824] | 3.33 [1.853 to 5.727]
  AngII at 24 hours: number analyzed (Participants) | 14 | 16
  AngII at 24 hours | 8.35 [4.506 to 15.378] | 2.41 [1.389 to 4.178]
  AngII at 48 hours: number analyzed (Participants) | 12 | 18
  AngII at 48 hours | 8.10 [4.219 to 15.071] | 3.74 [2.232 to 6.677]
  AngII at 48.5 hours: number analyzed (Participants) | 13 | 17
  AngII at 48.5 hours | 8.63 [4.514 to 15.961] | 2.89 [1.727 to 5.178]
  AngII at 50 hours: number analyzed (Participants) | 13 | 17
  AngII at 50 hours | 6.82 [3.551 to 12.510] | 2.58 [1.534 to 4.570]
  AngII at 54 hours: number analyzed (Participants) | 14 | 16
  AngII at 54 hours | 7.03 [3.770 to 12.850] | 2.32 [1.338 to 4.146]
  AngII at 60 hours: number analyzed (Participants) | 14 | 16
  AngII at 60 hours | 7.02 [3.883 to 12.768] | 2.38 [1.374 to 4.179]
  AngII at 66 hours: number analyzed (Participants) | 14 | 16
  AngII at 66 hours | 7.33 [4.156 to 13.262] | 1.84 [1.046 to 3.161]
  AngII at 72 hours: number analyzed (Participants) | 13 | 14
  AngII at 72 hours | 6.62 [3.701 to 12.174] | 1.93 [1.067 to 3.441]
  AngII at 96 hours: number analyzed (Participants) | 9 | 11
  AngII at 96 hours | 4.72 [2.325 to 9.769] | 1.70 [0.881 to 3.209]
  AngII at 120 hours: number analyzed (Participants) | 11 | 10
  AngII at 120 hours | 5.21 [3.036 to 10.126] | 2.64 [1.437 to 5.586]
  Ang1-5 at 0.5 hours: number analyzed (Participants) | 15 | 18
  Ang1-5 at 0.5 hours | 2.17 [1.408 to 3.376] | 8.58 [5.873 to 12.988]
  Ang1-5 at 2 hours: number analyzed (Participants) | 15 | 16
  Ang1-5 at 2 hours | 2.18 [1.410 to 3.383] | 7.50 [5.124 to 11.367]
  Ang1-5 at 6 hours: number analyzed (Participants) | 15 | 16
  Ang1-5 at 6 hours | 2.34 [1.508 to 3.643] | 8.38 [5.697 to 12.661]
  Ang1-5 at 12 hours: number analyzed (Participants) | 13 | 16
  Ang1-5 at 12 hours | 2.78 [1.784 to 4.363] | 5.07 [3.370 to 7.533]
  Ang1-5 at 24 hours: number analyzed (Participants) | 13 | 15
  Ang1-5 at 24 hours | 2.38 [1.512 to 3.763] | 3.57 [2.331 to 5.363]
  Ang1-5 at 48 hours: number analyzed (Participants) | 12 | 17
  Ang1-5 at 48 hours | 2.39 [1.519 to 3.724] | 4.59 [3.030 to 6.854]
  Ang1-5 at 48.5 hours: number analyzed (Participants) | 13 | 16
  Ang1-5 at 48.5 hours | 2.30 [1.465 to 3.568] | 5.26 [3.466 to 7.829]
  Ang1-5 at 50 hours: number analyzed (Participants) | 13 | 16
  Ang1-5 at 50 hours | 2.53 [1.619 to 3.924] | 4.91 [3.213 to 7.268]
  Ang1-5 at 54 hours: number analyzed (Participants) | 14 | 15
  Ang1-5 at 54 hours | 2.52 [1.629 to 3.936] | 3.21 [2.106 to 4.721]
  Ang1-5 at 60 hours: number analyzed (Participants) | 14 | 15
  Ang1-5 at 60 hours | 2.26 [1.478 to 3.490] | 2.78 [1.868 to 4.143]
  Ang1-5 at 66 hours: number analyzed (Participants) | 15 | 16
  Ang1-5 at 66 hours | 2.19 [1.454 to 3.366] | 2.71 [1.804 to 4.071]
  Ang1-5 at 72 hours: number analyzed (Participants) | 13 | 14
  Ang1-5 at 72 hours | 1.72 [1.125 to 2.662] | 2.50 [1.640 to 3.884]
  Ang1-5 at 96 hours: number analyzed (Participants) | 9 | 11
  Ang1-5 at 96 hours | 2.23 [1.315 to 3.822] | 1.28 [0.791 to 2.077]
  Ang1-5 at 120 hours: number analyzed (Participants) | 11 | 10
  Ang1-5 at 120 hours | 2.19 [1.451 to 3.412] | 1.38 [0.868 to 2.403]
  Ang1-7 at 0.5 hours: number analyzed (Participants) | 16 | 19
  Ang1-7 at 0.5 hours | 3.12 [1.702 to 5.665] | 13.15 [7.384 to 22.894]
  Ang1-7 at 2 hours: number analyzed (Participants) | 16 | 16
  Ang1-7 at 2 hours | 3.29 [1.786 to 5.965] | 12.05 [6.774 to 21.245]
  Ang1-7 at 6 hours: number analyzed (Participants) | 16 | 15
  Ang1-7 at 6 hours | 2.92 [1.578 to 5.361] | 15.33 [8.369 to 27.742]
  Ang1-7 at 12 hours: number analyzed (Participants) | 14 | 16
  Ang1-7 at 12 hours | 3.03 [1.607 to 5.711] | 6.82 [3.800 to 12.383]
  Ang1-7 at 24 hours: number analyzed (Participants) | 14 | 16
  Ang1-7 at 24 hours | 2.87 [1.514 to 5.410] | 6.25 [3.342 to 11.563]
  Ang1-7 at 48 hours: number analyzed (Participants) | 12 | 18
  Ang1-7 at 48 hours | 3.58 [1.878 to 6.875] | 5.71 [3.154 to 9.797]
  Ang1-7 at 48.5 hours: number analyzed (Participants) | 13 | 17
  Ang1-7 at 48.5 hours | 2.77 [1.472 to 5.289] | 5.54 [3.063 to 9.544]
  Ang1-7 at 50 hours: number analyzed (Participants) | 13 | 17
  Ang1-7 at 50 hours | 3.20 [1.696 to 6.064] | 6.13 [3.399 to 10.648]
  Ang1-7 at 54 hours: number analyzed (Participants) | 14 | 16
  Ang1-7 at 54 hours | 3.16 [1.686 to 6.031] | 5.78 [3.099 to 10.144]
  Ang1-7 at 60 hours: number analyzed (Participants) | 14 | 16
  Ang1-7 at 60 hours | 3.57 [1.907 to 6.701] | 4.74 [2.542 to 8.631]
  Ang1-7 at 66 hours: number analyzed (Participants) | 15 | 16
  Ang1-7 at 66 hours | 3.40 [1.837 to 6.298] | 3.97 [2.157 to 7.262]
  Ang1-7 at 72 hours: number analyzed (Participants) | 13 | 14
  Ang1-7 at 72 hours | 2.66 [1.389 to 5.051] | 4.70 [2.510 to 8.532]
  Ang1-7 at 96 hours: number analyzed (Participants) | 9 | 11
  Ang1-7 at 96 hours | 1.77 [0.796 to 3.823] | 2.43 [1.225 to 4.759]
  Ang1-7 at 120 hours: number analyzed (Participants) | 11 | 10
  Ang1-7 at 120 hours | 2.38 [1.213 to 4.155] | 3.21 [1.857 to 6.147]
Statistical Analysis 1: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); AngII, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 0.5 hours; Test type: Superiority or Other; p = 1.000, Bayesian repeated measures model; Ratio of Active/Placebo = 0.17, 95% CI 2-sided [0.083 to 0.359]
Statistical Analysis 2: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); AngII, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 2 hours; Test type: Superiority or Other; p = 0.9999, Bayesian repeated measures model; Ratio of Active/Placebo = 0.23, 95% CI 2-sided [0.111 to 0.492]
Statistical Analysis 3: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); AngII, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 6 hours; Test type: Superiority or Other; p = 0.9997, Bayesian repeated measures model; Ratio of Active/Placebo = 0.26, 95% CI 2-sided [0.121 to 0.568]
Statistical Analysis 4: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); AngII, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 12 hours; Test type: Superiority or Other; p = 0.9997, Bayesian repeated measures model; Ratio of Active/Placebo = 0.31, 95% CI 2-sided [0.136 to 0.660]
Statistical Analysis 5: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); AngII, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24 hours; Test type: Superiority or Other; p = 0.9991, Bayesian repeated measures model; Ratio of Active/Placebo = 0.29, 95% CI 2-sided [0.133 to 0.632]
Statistical Analysis 6: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); AngII, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48 hours; Test type: Superiority or Other; p = 0.9631, Bayesian repeated measures model; Ratio of Active/Placebo = 0.46, 95% CI 2-sided [0.213 to 1.081]
Statistical Analysis 7: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); AngII, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48.5 hours; Test type: Superiority or Other; p = 0.9941, Bayesian repeated measures model; Ratio of Active/Placebo = 0.33, 95% CI [0.157 to 0.789]
Statistical Analysis 8: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); AngII, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 50 hours; Test type: Superiority or Other; p = 0.9875, Bayesian repeated measures model; Ratio of Active/Placebo = 0.38, 95% CI 2-sided [0.179 to 0.891]
Statistical Analysis 9: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); AngII, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 54 hours; Test type: Superiority or Other; p = 0.9956, Bayesian repeated measures model; Ratio of Active/Placebo = 0.33, 95% CI 2-sided [0.151 to 0.759]
Statistical Analysis 10: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); AngII, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 60 hours; Test type: Superiority or Other; p = 0.9964, Bayesian repeated measures model; Ratio of Active/Placebo = 0.34, 95% CI 2-sided [0.157 to 0.747]
Statistical Analysis 11: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); AngII, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 66 hours; Test type: Superiority or Other; p = 0.9999, Bayesian repeated measures model; Ratio of Active/Placebo = 0.25, 95% CI 2-sided [0.114 to 0.532]
Statistical Analysis 12: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); AngII, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority or Other; p = 0.9991, Bayesian repeated measures model; Ratio of Active/Placebo = 0.29, 95% CI 2-sided [0.130 to 0.647]
Statistical Analysis 13: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); AngII, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 96 hours; Test type: Superiority or Other; p = 0.9852, Bayesian repeated measures model; Ratio of Active/Placebo = 0.36, 0.9852% CI 2-sided [0.137 to 0.906]
Statistical Analysis 14: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); AngII, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 120 hours; Test type: Superiority or Other; p = 0.9719, Bayesian repeated measures model; Ratio of Active/Placebo = 0.51, 95% CI 2-sided [0.230 to 1.014]
Statistical Analysis 15: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-5 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 0.5 hours; Test type: Superiority; p = 1.0000, Bayesian repeated measures model; Ratio of Active/Placebo = 3.98, 95% CI 2-sided [2.263 to 6.919]
Statistical Analysis 16: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-5 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 2 hours; Test type: Superiority or Other; p = 1.000, Bayesian repeated measures model; Ratio of Active/Placebo = 3.46, 95% CI 2-sided [1.976 to 6.052]
Statistical Analysis 17: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-5 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 6 hours; Test type: Superiority or Other; p = 1.0000, Bayesian repeated measures model; Ratio of Active/Placebo = 3.59, 95% CI 2-sided [2.060 to 6.345]
Statistical Analysis 18: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-5 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 12 hours; Test type: Superiority or Other; p = 0.9806, Bayesian repeated measures model; Ratio of Active/Placebo = 1.82, 95% CI 2-sided [1.031 to 3.170]
Statistical Analysis 19: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-5 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24 hours; Test type: Superiority; p = 0.9129, Bayesian repeated measures model; Ratio of Active/Placebo = 1.50, 95% CI 2-sided [0.828 to 2.636]
Statistical Analysis 20: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-5 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48 hours; Test type: Superiority; p = 0.9891, Bayesian repeated measures model; Ratio of Active/Placebo = 1.92, 95% CI 2-sided [1.098 to 3.349]
Statistical Analysis 21: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-5 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48.5 hours; Test type: Superiority or Other; p = 0.9983, Bayesian repeated measures model; Ratio of Active/Placebo = 2.29, 95% CI 2-sided [1.316 to 3.974]
Statistical Analysis 22: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-5 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 50 hours; Test type: Superiority or Other; p = 0.9900, Bayesian repeated measures model; Ratio of Active/Placebo = 1.94, 95% CI 2-sided [1.112 to 3.359]
Statistical Analysis 23: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-5 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 54 hours; Test type: Superiority or Other; p = 0.7996, Bayesian repeated measures model; Ratio of Active/Placebo = 1.27, 95% CI 2-sided [0.729 to 2.163]
Statistical Analysis 24: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-5 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 60 hours; Test type: Superiority or Other; p = 0.7778, Bayesian repeated measures model; Ratio of Active/Placebo = 1.23, 95% CI 2-sided [0.718 to 2.087]
Statistical Analysis 25: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-5 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 66 hours; Test type: Superiority or Other; p = 0.7730, Bayesian repeated measures model; Ratio of Active/Placebo = 1.24, 95% CI 2-sided [0.705 to 2.113]
Statistical Analysis 26: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-5 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority or Other; p = 0.8951, Bayesian repeated measures model; Ratio of Active/Placebo = 1.45, 95% CI 2-sided [0.814 to 2.604]
Statistical Analysis 27: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-5 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 96 hours; Test type: Superiority or Other; p = 0.9324, Bayesian repeated measures model; Ratio of Active/Placebo = 0.57, 95% CI 2-sided [0.276 to 1.183]
Statistical Analysis 28: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-5 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 120 hours; Test type: Superiority or Other; p = 0.8982, Bayesian repeated measures model; Ratio of Active/Placebo = 0.63, 95% CI 2-sided [0.351 to 1.257]
Statistical Analysis 29: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-7 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 0.5 hours; Test type: Superiority or Other; p = 0.9998, Bayesian repeated measures model; Ratio of Active/Placebo = 4.22, 95% CI 2-sided [1.910 to 8.905]
Statistical Analysis 30: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-7 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 2 hours; Test type: Superiority or Other; p = 0.9993, Bayesian repeated measures model; Ratio of Active/Placebo = 3.67, 95% CI 2-sided [1.689 to 7.970]
Statistical Analysis 31: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-7 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 6 hours; Test type: Superiority or Other; p = 1.0000, Bayesian repeated measures model; Ratio of Active/Placebo = 5.26, 95% CI 2-sided [2.392 to 11.754]
Statistical Analysis 32: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-7 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 12 hours; Test type: Superiority or Other; p = 0.9713, Bayesian repeated measures model; Ratio of Active/Placebo = 2.25, 95% CI 2-sided [0.972 to 5.136]
Statistical Analysis 33: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-7 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24 hours; Test type: Superiority or Other; p = 0.9649, Bayesian repeated measures model; Ratio of Active/Placebo = 2.19, 95% CI 2-sided [0.940 to 4.975]
Statistical Analysis 34: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-7 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48 hours; Test type: Superiority or Other; p = 0.8749, Mixed Models Analysis; Ratio of Active/Placebo = 1.59, 95% CI 2-sided [0.711 to 3.473]
Statistical Analysis 35: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-7 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48.5 hours; Test type: Superiority or Other; p = 0.9566, Bayesian repeated measures model; Ratio of Active/Placebo = 1.99, 95% CI 2-sided [0.899 to 4.342]
Statistical Analysis 36: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-7 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 50 hours; Test type: Superiority or Other; p = 0.9549, Bayesian repeated measures model; Ratio of Active/Placebo = 1.91, 95% CI 2-sided [0.862 to 4.173]
Statistical Analysis 37: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-7 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 54 hours; Test type: Superiority or Other; p = 0.9275, Bayesian repeated measures model; Ratio of Active/Placebo = 1.81, 95% CI 2-sided [0.816 to 4.005]
Statistical Analysis 38: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-7 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 60 hours; Test type: Superiority; p = 0.7483, Bayesian repeated measures model; Ratio of Active/Placebo = 1.32, 95% CI 2-sided [0.584 to 3.007]
Statistical Analysis 39: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-7 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 66 hours; Test type: Superiority or Other; p = 0.6480, Bayesian repeated measures model; Ratio of Active/Placebo = 1.17, 95% CI 2-sided [0.516 to 2.675]
Statistical Analysis 40: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-7 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority or Other; p = 0.9038, Bayesian repeated measures model; Ratio of Active/Placebo = 1.76, 95% CI 2-sided [0.741 to 4.170]
Statistical Analysis 41: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-7 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 96 hours; Test type: Superiority or Other; p = 0.7339, Bayesian repeated measures model; Ratio of Active/Placebo = 1.38, 95% CI 2-sided [0.490 to 3.915]
Statistical Analysis 42: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang1-7 , Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 120 hours; Test type: Superiority or Other; p = 0.7714, Bayesian repeated measures model; Ratio of Active/Placebo = 1.38, 95% CI 2-sided [0.651 to 3.321]

23. Secondary Outcome: Pharmacodynamic/Biomarker Analysis (Renin-angiotensin System Cascade Biomarkers) to Include Ang II/Ang (1-5) and Ang II/Ang (1-7) Upto Day 5(Part B)
Description: Renin-angiotensin system cascade biomarkers included Ang II/Ang (1-5) and Ang II/Ang (1-7) and). Blood samples for biomarker analyses were collected 0.5 hours, 2 hours, 6 hours, 12 hours, 24 hours, 48 hours, 48.5 hours, 50 hours, 54 hours, 60 hours, 66 hours, 72 hours, 96 hours and 120 hours upto Day 5. Data has been presented for median along with the 95% credible interval.
Time Frame: as for outcome 22
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Median (95% Confidence Interval); unit: Ratio
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
Ratio
  Ang II/Ang1-5 at 0.5 hours: number analyzed (Participants) | 16 | 18
  Ang II/Ang1-5 at 0.5 hours | 4.35 [2.463 to 7.664] | 0.29 [0.175 to 0.488]
  Ang II/Ang1-5 at 2 hours: number analyzed (Participants) | 16 | 16
  Ang II/Ang1-5 at 2 hours | 3.82 [2.150 to 6.713] | 0.38 [0.227 to 0.645]
  Ang II/Ang1-5 at 6 hours: number analyzed (Participants) | 16 | 15
  Ang II/Ang1-5 at 6 hours | 3.20 [1.793 to 5.619] | 0.36 [0.211 to 0.629]
  Ang II/Ang1-5 at 12 hours: number analyzed (Participants) | 14 | 15
  Ang II/Ang1-5 at 12 hours | 2.90 [1.605 to 5.215] | 0.72 [0.414 to 1.270]
  Ang II/Ang1-5 at 24 hours: number analyzed (Participants) | 14 | 15
  Ang II/Ang1-5 at 24 hours | 2.35 [1.296 to 4.276] | 0.68 [0.383 to 1.182]
  Ang II/Ang1-5 at 48 hours: number analyzed (Participants) | 13 | 17
  Ang II/Ang1-5 at 48 hours | 2.68 [1.481 to 4.757] | 0.85 [0.497 to 1.445]
  Ang II/Ang1-5 at 48.5 hours: number analyzed (Participants) | 14 | 16
  Ang II/Ang1-5 at 48.5 hours | 2.90 [1.606 to 5.164] | 0.56 [0.328 to 0.959]
  Ang II/Ang1-5 at 50 hours: number analyzed (Participants) | 14 | 16
  Ang II/Ang1-5 at 50 hours | 2.11 [1.181 to 3.740] | 0.53 [0.311 to 0.909]
  Ang II/Ang1-5 at 54 hours: number analyzed (Participants) | 15 | 15
  Ang II/Ang1-5 at 54 hours | 2.21 [1.249 to 3.885] | 0.68 [0.385 to 1.191]
  Ang II/Ang1-5 at 60 hours: number analyzed (Participants) | 15 | 15
  Ang II/Ang1-5 at 60 hours | 2.52 [1.445 to 4.412] | 0.86 [0.496 to 1.501]
  Ang II/Ang1-5 at 66 hours: number analyzed (Participants) | 15 | 16
  Ang II/Ang1-5 at 66 hours | 2.90 [1.669 to 5.036] | 0.64 [0.370 to 1.105]
  Ang II/Ang1-5 at 72 hours: number analyzed (Participants) | 14 | 14
  Ang II/Ang1-5 at 72 hours | 2.91 [1.620 to 5.153] | 0.76 [0.429 to 1.335]
  Ang II/Ang1-5 at 96 hours: number analyzed (Participants) | 10 | 11
  Ang II/Ang1-5 at 96 hours | 1.72 [0.870 to 3.387] | 1.41 [0.738 to 2.695]
  Ang II/Ang1-5 at 120 hours: number analyzed (Participants) | 12 | 10
  Ang II/Ang1-5 at 120 hours | 1.93 [1.058 to 3.508] | 1.53 [0.768 to 2.872]
  Ang II/Ang1-7 at 0.5 hours: number analyzed (Participants) | 17 | 18
  Ang II/Ang1-7 at 0.5 hours | 3.10 [1.681 to 5.669] | 0.19 [0.110 to 0.342]
  Ang II/Ang1-7 at 2 hours: number analyzed (Participants) | 17 | 16
  Ang II/Ang1-7 at 2 hours | 2.52 [1.379 to 4.611] | 0.24 [0.135 to 0.432]
  Ang II/Ang1-7 at 6 hours: number analyzed (Participants) | 17 | 14
  Ang II/Ang1-7 at 6 hours | 2.63 [1.456 to 4.767] | 0.20 [0.109 to 0.378]
  Ang II/Ang1-7 at 12 hours: number analyzed (Participants) | 15 | 15
  Ang II/Ang1-7 at 12 hours | 2.50 [1.352 to 4.675] | 0.49 [0.267 to 0.913]
  Ang II/Ang1-7 at 24 hours: number analyzed (Participants) | 15 | 16
  Ang II/Ang1-7 at 24 hours | 2.11 [1.127 to 3.990] | 0.37 [0.200 to 0.671]
  Ang II/Ang1-7 at 48 hours: number analyzed (Participants) | 13 | 18
  Ang II/Ang1-7 at 48 hours | 1.61 [0.843 to 3.105] | 0.65 [0.363 to 1.146]
  Ang II/Ang1-7 at 48.5 hours: number analyzed (Participants) | 14 | 17
  Ang II/Ang1-7 at 48.5 hours | 2.18 [1.147 to 4.165] | 0.51 [0.291 to 0.917]
  Ang II/Ang1-7 at 50 hours: number analyzed (Participants) | 14 | 17
  Ang II/Ang1-7 at 50 hours | 1.51 [0.799 to 2.887] | 0.42 [0.233 to 0.747]
  Row 23Ang II/Ang1-7 at 54 hours: number analyzed (Participants) | 15 | 16
  Row 23Ang II/Ang1-7 at 54 hours | 1.64 [0.872 to 3.105] | 0.40 [0.213 to 0.719]
  Ang II/Ang1-7 at 60 hours: number analyzed (Participants) | 15 | 16
  Ang II/Ang1-7 at 60 hours | 1.55 [0.817 to 2.945] | 0.48 [0.264 to 0.878]
  Ang II/Ang1-7 at 66 hours: number analyzed (Participants) | 15 | 16
  Ang II/Ang1-7 at 66 hours | 1.81 [0.964 to 3.354] | 0.45 [0.246 to 0.825]
  Ang II/Ang1-7 at 72 hours: number analyzed (Participants) | 14 | 14
  Ang II/Ang1-7 at 72 hours | 1.75 [0.931 to 3.295] | 0.42 [0.219 to 0.796]
  Ang II/Ang1-7 at 96 hours: number analyzed (Participants) | 10 | 11
  Ang II/Ang1-7 at 96 hours | 2.02 [0.951 to 4.323] | 0.69 [0.335 to 1.406]
  Ang II/Ang1-7 at 120 hours: number analyzed (Participants) | 12 | 10
  Ang II/Ang1-7 at 120 hours | 1.66 [0.826 to 3.178] | 0.64 [0.311 to 1.568]
Statistical Analysis 1: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-5, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 0.5 hours; Test type: Superiority or Other; p = 1.0000, Bayesian repeated measures model; Ratio of Active/Placebo = 0.07, 95% CI 2-sided [0.032 to 0.140]
Statistical Analysis 2: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-5, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 2 hours; Test type: Superiority or Other; p = 1.0000, Bayesian repeated measures model; Ratio of Active/Placebo = 0.10, 95% CI 2-sided [0.048 to 0.209]
Statistical Analysis 3: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-5, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 6 hours; Test type: Superiority or Other; p = 1.0000, Bayesian repeated measures model; Ratio of Active/Placebo = 0.11, 95% CI 2-sided [0.054 to 0.243]
Statistical Analysis 4: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-5, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 12 hours; Test type: Superiority or Other; p = 0.9996, Bayesian repeated measures model; Ratio of Active/Placebo = 0.25, 95% CI 2-sided [0.113 to 0.547]
Statistical Analysis 5: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-5, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24 hours; Test type: Superiority or Other; p = 0.9991, Bayesian repeated measures model; Ratio of Active/Placebo = 0.29, 95% CI 2-sided [0.130 to 0.634]
Statistical Analysis 6: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-5, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48 hours; Test type: Superiority or Other; p = 0.9979, Bayesian repeated measures model; Ratio of Active/Placebo = 0.32, 95% CI 2-sided [0.149 to 0.682]
Statistical Analysis 7: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-5, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48.5 hours; Test type: Superiority or Other; p = 1.0000, Bayesian repeated measures model; Ratio of Active/Placebo = 0.19, 95% CI [0.091 to 0.417]
Statistical Analysis 8: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-5, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 50 hours; Test type: Superiority or Other; p = 0.9998, Bayesian repeated measures model; Ratio of Active/Placebo = 0.25, 95% CI 2-sided [0.119 to 0.539]
Statistical Analysis 9: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-5, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 54 hours; Test type: Superiority or Other; p = 0.9985, Bayesian repeated measures model; Ratio of Active/Placebo = 0.31, 95% CI 2-sided [0.141 to 0.666]
Statistical Analysis 10: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-5, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 60 hours; Test type: Superiority or Other; p = 0.9977, Bayesian repeated measures model; Ratio of Active/Placebo = 0.34, 95% CI 2-sided [0.162 to 0.730]
Statistical Analysis 11: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-5, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 66 hours; Test type: Superiority or Other; p = 0.9999, Bayesian repeated measures model; Ratio of Active/Placebo = 0.22, 95% CI 2-sided [0.105 to 0.468]
Statistical Analysis 12: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-5, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority or Other; p = 0.9996, Bayesian repeated measures model; Ratio of Active/Placebo = 0.26, 95% CI 2-sided [0.119 to 0.570]
Statistical Analysis 13: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-5, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 96 hours; Test type: Superiority or Other; p = 0.6621, Bayesian repeated measures model; Ratio of Active/Placebo = 0.82, 95% CI 2-sided [0.319 to 2.136]
Statistical Analysis 14: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-5, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 120 hours; Test type: Superiority or Other; p = 0.7085, Bayesian repeated measures model; Ratio of Active/Placebo = 0.79, 95% CI 2-sided [0.324 to 1.847]
Statistical Analysis 15: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-7, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 0.5 hours; Test type: Superiority or Other; p = 1.0000, Bayesian repeated measures model; Ratio of Active/Placebo = 0.06, 95% CI 2-sided [0.028 to 0.140]
Statistical Analysis 16: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-7, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 2 hours; Test type: Superiority or Other; p = 1.0000, Bayesian repeated measures model; Ratio of Active/Placebo = 0.10, 95% CI 2-sided [0.043 to 0.216]
Statistical Analysis 17: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-7, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 6 hours; Test type: Superiority or Other; p = 1.0000, Bayesian repeated measures model; Ratio of Active/Placebo = 0.08, 95% CI 2-sided [0.034 to 0.177]
Statistical Analysis 18: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-7, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 12 hours; Test type: Superiority or Other; p = 0.9998, Bayesian repeated measures model; Ratio of Active/Placebo = 0.20, 95% CI 2-sided [0.086 to 0.453]
Statistical Analysis 19: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-7, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24 hours; Test type: Superiority or Other; p = 0.9999, Bayesian repeated measures model; Ratio of Active/Placebo = 0.17, 95% CI 2-sided [0.075 to 0.400]
Statistical Analysis 20: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-7, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48 hours; Test type: Superiority or Other; p = 0.9863, Bayesian repeated measures model; Ratio of Active/Placebo = 0.40, 95% CI 2-sided [0.173 to 0.901]
Statistical Analysis 21: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-7, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48.5 hours; Test type: Superiority or Other; p = 0.9998, Bayesian repeated measures model; Ratio of Active/Placebo = 0.24, 95% CI 2-sided [0.103 to 0.529]
Statistical Analysis 22: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-7, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 50 hours; Test type: Superiority or Other; p = 0.9992, Bayesian repeated measures model; Ratio of Active/Placebo = 0.28, 95% CI 2-sided [0.119 to 0.626]
Statistical Analysis 23: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-7, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 54 hours; Test type: Superiority or Other; p = 0.9995, Bayesian repeated measures model; Ratio of Active/Placebo = 0.24, 95% CI 2-sided [0.102 to 0.561]
Statistical Analysis 24: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-7, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 60 hours; Test type: Superiority or Other; p = 0.9964, Bayesian repeated measures model; Ratio of Active/Placebo = 0.31, 95% CI 2-sided [0.131 to 0.729]
Statistical Analysis 25: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-7, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 66 hours; Test type: Superiority or Other; p = 0.9995, Bayesian repeated measures model; Ratio of Active/Placebo = 0.25, 95% CI 2-sided [0.107 to 0.584]
Statistical Analysis 26: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-7, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority or Other; p = 0.9993, Ratio of Active/Placebo; Ratio of Active/Placebo = 0.24, 95% CI 2-sided [0.098 to 0.578]
Statistical Analysis 27: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-7, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 96 hours; Test type: Superiority or Other; p = 0.9781, Bayesian repeated measures model; Ratio of Active/Placebo = 0.34, 95% CI 2-sided [0.119 to 0.969]
Statistical Analysis 28: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Ang II/Ang1-7, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 120 hours; Test type: Superiority or Other; p = 0.9375, Bayesian repeated measures model; Ratio of Active/Placebo = 0.38, 95% CI 2-sided [0.154 to 1.341]

24. Secondary Outcome: Measures of Oxygenation Including Level of Positive End Expiratory Pressure (PEEP), Peak Ventilatory Pressures and Plateau Ventilatory Pressures Upto Day 7 (Part B)
Description: Measures of oxygenation included PEEP the pressure in the lungs (alveolar pressure) above atmospheric pressure (the pressure outside of the body) that exists at the end of expiration, peak ventilator pressure highest level of pressure applied to the lungs during inhalation and plateau ventilatory pressure the pressure applied to small airways and alveoli measured during an inspiratory pause on the ventilator. Assessments were performed at 0.5, 1, 2, 4, 6, 8, 12, 18, 24, 24.5, 25, 26, 28, 30, 32, 36, 42, 48, 48.5, 49, 50, 52, 54, 56, 60, 66, 72 and 168 hours upto Day 7. Data has been presented for median along with the 95% credible interval.
Time Frame: 0.5, 1, 2, 4, 6, 8, 12, 18, 24, 24.5, 25, 26, 28, 30, 32, 36, 42, 48, 48.5, 49, 50, 52, 54, 56, 60, 66, 72 and 168 hours upto Day 7
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Median (90% Confidence Interval); unit: centimeters of water pressure
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
centimeters of water pressure
  PEEP at 0.5 hours: number analyzed (Participants) | 16 | 18
  PEEP at 0.5 hours | 10.3 [8.87 to 12.18] | 9.6 [8.23 to 11.54]
  PEEP at 1 hour: number analyzed (Participants) | 17 | 18
  PEEP at 1 hour | 9.9 [8.51 to 11.69] | 9.6 [8.23 to 11.60]
  PEEP at 2 hours: number analyzed (Participants) | 16 | 17
  PEEP at 2 hours | 9.9 [8.48 to 11.62] | 9.7 [8.26 to 11.72]
  PEEP at 4 hours: number analyzed (Participants) | 17 | 18
  PEEP at 4 hours | 9.7 [8.30 to 11.29] | 9.6 [8.21 to 11.56]
  PEEP at 6 hours: number analyzed (Participants) | 16 | 18
  PEEP at 6 hours | 9.6 [8.28 to 11.14] | 9.5 [8.21 to 11.32]
  PEEP at 8 hours: number analyzed (Participants) | 17 | 17
  PEEP at 8 hours | 9.7 [8.38 to 11.18] | 9.6 [8.25 to 11.19]
  PEEP at 12 hours: number analyzed (Participants) | 15 | 18
  PEEP at 12 hours | 9.8 [8.56 to 11.38] | 9.5 [8.13 to 10.87]
  PEEP at 18 hours: number analyzed (Participants) | 17 | 18
  PEEP at 18 hours | 10.1 [8.79 to 11.71] | 9.6 [8.23 to 11.13]
  PEEP at 24 hours: number analyzed (Participants) | 16 | 18
  PEEP at 24 hours | 9.7 [8.39 to 11.36] | 9.3 [8.13 to 10.76]
  PEEP at 24.5 hours: number analyzed (Participants) | 16 | 17
  PEEP at 24.5 hours | 9.7 [8.39 to 11.37] | 9.3 [8.14 to 10.78]
  PEEP at 25 hours: number analyzed (Participants) | 16 | 18
  PEEP at 25 hours | 9.7 [8.41 to 11.38] | 8.6 [7.47 to 9.89]
  PEEP at 26 hours: number analyzed (Participants) | 16 | 17
  PEEP at 26 hours | 9.4 [8.13 to 11.01] | 9.3 [8.11 to 10.78]
  PEEP at 28 hours: number analyzed (Participants) | 16 | 17
  PEEP at 28 hours | 9.1 [7.89 to 10.70] | 9.4 [8.02 to 10.79]
  PEEP at 30 hours: number analyzed (Participants) | 15 | 18
  PEEP at 30 hours | 9.5 [8.20 to 11.11] | 9.3 [7.89 to 10.78]
  PEEP at 32 hours: number analyzed (Participants) | 15 | 18
  PEEP at 32 hours | 9.1 [7.84 to 10.63] | 9.2 [7.79 to 10.66]
  PEEP at 36 hours: number analyzed (Participants) | 14 | 18
  PEEP at 36 hours | 9.3 [7.91 to 10.96] | 9.0 [7.75 to 10.55]
  PEEP at 42 hours: number analyzed (Participants) | 15 | 18
  PEEP at 42 hours | 9.6 [8.21 to 11.31] | 8.9 [7.59 to 10.39]
  PEEP at 48 hours: number analyzed (Participants) | 14 | 16
  PEEP at 48 hours | 9.6 [8.20 to 11.38] | 8.8 [7.52 to 10.40]
  PEEP at 48.5 hours: number analyzed (Participants) | 13 | 17
  PEEP at 48.5 hours | 9.6 [8.19 to 11.42] | 8.8 [7.57 to 10.47]
  PEEP at 49 hours: number analyzed (Participants) | 13 | 17
  PEEP at 49 hours | 9.6 [8.17 to 11.44] | 8.6 [7.43 to 10.26]
  PEEP at 50 hours: number analyzed (Participants) | 13 | 17
  PEEP at 50 hours | 9.6 [8.12 to 11.39] | 8.7 [7.50 to 10.34]
  PEEP at 52 hours: number analyzed (Participants) | 13 | 16
  PEEP at 52 hours | 9.6 [8.18 to 11.48] | 8.8 [7.56 to 10.45]
  PEEP at 54 hours: number analyzed (Participants) | 14 | 17
  PEEP at 54 hours | 9.4 [7.98 to 11.25] | 8.7 [7.41 to 10.19]
  PEEP at 56 hours: number analyzed (Participants) | 13 | 16
  PEEP at 56 hours | 9.2 [7.85 to 11.12] | 8.7 [7.38 to 10.16]
  PEEP at 60 hours: number analyzed (Participants) | 13 | 15
  PEEP at 60 hours | 8.9 [7.55 to 10.62] | 8.2 [6.91 to 9.63]
  PEEP at 66 hours: number analyzed (Participants) | 11 | 13
  PEEP at 66 hours | 9.4 [7.85 to 11.04] | 9.1 [7.56 to 10.63]
  PEEP at 72 hours: number analyzed (Participants) | 11 | 13
  PEEP at 72 hours | 9.6 [7.98 to 11.34] | 8.8 [7.53 to 10.25]
  PEEP at 168 hours: number analyzed (Participants) | 4 | 7
  PEEP at 168 hours | 6.9 [5.83 to 9.05] | 7.5 [6.19 to 9.36]
  Peak ventilatory pressure at 0.5 hours: number analyzed (Participants) | 17 | 16
  Peak ventilatory pressure at 0.5 hours | 29.3 [26.72 to 32.02] | 29.7 [27.00 to 32.70]
  Peak ventilatory pressure at 1 hour: number analyzed (Participants) | 16 | 16
  Peak ventilatory pressure at 1 hour | 28.3 [25.83 to 30.98] | 30.4 [27.58 to 33.38]
  Peak ventilatory pressure at 2 hours: number analyzed (Participants) | 16 | 16
  Peak ventilatory pressure at 2 hours | 27.7 [25.37 to 30.43] | 29.7 [26.78 to 32.67]
  Peak ventilatory pressure at 4 hours: number analyzed (Participants) | 15 | 16
  Peak ventilatory pressure at 4 hours | 28.4 [25.94 to 31.06] | 28.8 [25.99 to 31.64]
  Peak ventilatory pressure at 6 hours: number analyzed (Participants) | 17 | 16
  Peak ventilatory pressure at 6 hours | 28.1 [25.77 to 30.74] | 29.4 [26.63 to 32.33]
  Peak ventilatory pressure at 8 hours: number analyzed (Participants) | 16 | 16
  Peak ventilatory pressure at 8 hours | 28.2 [25.78 to 30.91] | 29.3 [26.48 to 32.15]
  Peak ventilatory pressure at 12 hours: number analyzed (Participants) | 16 | 16
  Peak ventilatory pressure at 12 hours | 28.5 [25.94 to 31.18] | 29.7 [27.04 to 32.59]
  Peak ventilatory pressure at 18 hours: number analyzed (Participants) | 16 | 15
  Peak ventilatory pressure at 18 hours | 29.5 [26.87 to 32.31] | 28.9 [26.21 to 31.79]
  Peak ventilatory pressure at 24 hours: number analyzed (Participants) | 16 | 16
  Peak ventilatory pressure at 24 hours | 28.8 [26.30 to 31.56] | 28.3 [25.66 to 31.08]
  Peak ventilatory pressure at 24.5 hours: number analyzed (Participants) | 16 | 15
  Peak ventilatory pressure at 24.5 hours | 29.1 [26.61 to 31.96] | 28.2 [25.66 to 31.04]
  Peak ventilatory pressure at 25 hours: number analyzed (Participants) | 16 | 16
  Peak ventilatory pressure at 25 hours | 29.4 [26.80 to 32.24] | 27.2 [24.74 to 29.92]
  Peak ventilatory pressure at 26 hours: number analyzed (Participants) | 15 | 15
  Peak ventilatory pressure at 26 hours | 27.6 [25.10 to 30.26] | 27.4 [24.87 to 30.15]
  Peak ventilatory pressure at 28 hours: number analyzed (Participants) | 16 | 14
  Peak ventilatory pressure at 28 hours | 29.3 [26.64 to 32.27] | 26.9 [24.32 to 29.57]
  Peak ventilatory pressure at 30 hours: number analyzed (Participants) | 15 | 16
  Peak ventilatory pressure at 30 hours | 29.5 [26.81 to 32.52] | 28.6 [26.00 to 31.36]
  Peak ventilatory pressure at 32 hours: number analyzed (Participants) | 16 | 15
  Peak ventilatory pressure at 32 hours | 30.7 [27.98 to 33.72] | 28.1 [25.44 to 30.81]
  Peak ventilatory pressure at 36 hours: number analyzed (Participants) | 15 | 15
  Peak ventilatory pressure at 36 hours | 30.7 [27.79 to 33.74] | 27.0 [24.29 to 29.68]
  Peak ventilatory pressure at 42 hours: number analyzed (Participants) | 14 | 16
  Peak ventilatory pressure at 42 hours | 28.2 [25.52 to 31.26] | 27.6 [25.01 to 30.23]
  Peak ventilatory pressure at 48 hours: number analyzed (Participants) | 14 | 13
  Peak ventilatory pressure at 48 hours | 25.7 [23.17 to 28.40] | 26.7 [24.13 to 29.47]
  Peak ventilatory pressure at 48.5 hours: number analyzed (Participants) | 13 | 13
  Peak ventilatory pressure at 48.5 hours | 26.0 [23.41 to 28.78] | 28.1 [25.40 to 31.03]
  Peak ventilatory pressure at 49 hours: number analyzed (Participants) | 13 | 13
  Peak ventilatory pressure at 49 hours | 26.4 [23.71 to 29.23] | 28.1 [25.34 to 30.97]
  Peak ventilatory pressure at 50 hours: number analyzed (Participants) | 13 | 13
  Peak ventilatory pressure at 50 hours | 24.2 [21.79 to 26.86] | 27.3 [24.59 to 30.19]
  Peak ventilatory pressure at 52 hours: number analyzed (Participants) | 12 | 12
  Peak ventilatory pressure at 52 hours | 26.6 [23.87 to 29.57] | 26.7 [24.12 to 29.47]
  Peak ventilatory pressure at 54 hours: number analyzed (Participants) | 14 | 13
  Peak ventilatory pressure at 54 hours | 25.3 [22.87 to 27.95] | 27.3 [24.76 to 30.15]
  Peak ventilatory pressure at 56 hours: number analyzed (Participants) | 12 | 12
  Peak ventilatory pressure at 56 hours | 25.6 [23.14 to 28.43] | 27.9 [25.22 to 31.07]
  Peak ventilatory pressure at 60 hours: number analyzed (Participants) | 13 | 12
  Peak ventilatory pressure at 60 hours | 24.1 [21.79 to 26.75] | 26.8 [24.09 to 29.82]
  Peak ventilatory pressure at 66 hours: number analyzed (Participants) | 10 | 11
  Peak ventilatory pressure at 66 hours | 24.3 [21.48 to 27.38] | 25.9 [23.08 to 28.92]
  Peak ventilatory pressure at 72 hours: number analyzed (Participants) | 7 | 9
  Peak ventilatory pressure at 72 hours | 22.9 [20.08 to 26.34] | 29.3 [25.85 to 32.87]
  Peak ventilatory pressure at 168 hours: number analyzed (Participants) | 3 | 5
  Peak ventilatory pressure at 168 hours | 19.9 [17.35 to 24.63] | 25.2 [20.70 to 30.23]
  Plateau ventilatory pressure at 0.5 hours: number analyzed (Participants) | 10 | 12
  Plateau ventilatory pressure at 0.5 hours | 24.2 [21.41 to 27.12] | 25.9 [23.02 to 29.17]
  Plateau ventilatory pressure at 1 hour: number analyzed (Participants) | 12 | 12
  Plateau ventilatory pressure at 1 hour | 24.8 [22.06 to 27.85] | 24.7 [21.90 to 27.72]
  Plateau ventilatory pressure at 2 hours: number analyzed (Participants) | 9 | 11
  Plateau ventilatory pressure at 2 hours | 23.9 [21.22 to 26.96] | 24.8 [21.92 to 27.89]
  Plateau ventilatory pressure at 4 hours: number analyzed (Participants) | 9 | 10
  Plateau ventilatory pressure at 4 hours | 24.3 [21.65 to 27.49] | 24.9 [21.95 to 28.22]
  Plateau ventilatory pressure at 6 hours: number analyzed (Participants) | 12 | 10
  Plateau ventilatory pressure at 6 hours | 24.8 [22.15 to 27.77] | 25.2 [22.07 to 28.62]
  Plateau ventilatory pressure at 8 hours: number analyzed (Participants) | 13 | 10
  Plateau ventilatory pressure at 8 hours | 25.9 [23.20 to 29.05] | 21.9 [19.22 to 24.84]
  Plateau ventilatory pressure at 12 hours: number analyzed (Participants) | 11 | 10
  Plateau ventilatory pressure at 12 hours | 24.1 [21.38 to 27.26] | 24.0 [20.96 to 27.38]
  Plateau ventilatory pressure at 18 hours: number analyzed (Participants) | 11 | 8
  Plateau ventilatory pressure at 18 hours | 25.3 [22.45 to 28.64] | 21.5 [18.63 to 24.95]
  Plateau ventilatory pressure at 24 hours: number analyzed (Participants) | 10 | 10
  Plateau ventilatory pressure at 24 hours | 24.1 [21.46 to 27.25] | 24.2 [21.16 to 27.44]
  Plateau ventilatory pressure at 24.5 hours: number analyzed (Participants) | 11 | 10
  Plateau ventilatory pressure at 24.5 hours | 23.8 [21.22 to 26.84] | 23.2 [20.36 to 26.37]
  Plateau ventilatory pressure at 25 hours: number analyzed (Participants) | 11 | 9
  Plateau ventilatory pressure at 25 hours | 24.4 [21.74 to 27.49] | 22.2 [19.44 to 25.35]
  Plateau ventilatory pressure at 26 hours: number analyzed (Participants) | 9 | 10
  Plateau ventilatory pressure at 26 hours | 23.3 [20.70 to 26.42] | 23.2 [20.26 to 26.72]
  Plateau ventilatory pressure at 28 hours: number analyzed (Participants) | 11 | 10
  Plateau ventilatory pressure at 28 hours | 23.1 [20.47 to 26.03] | 23.4 [20.43 to 26.90]
  Plateau ventilatory pressure at 30 hours: number analyzed (Participants) | 9 | 10
  Plateau ventilatory pressure at 30 hours | 23.3 [20.44 to 26.61] | 23.6 [20.71 to 27.01]
  Plateau ventilatory pressure at 32 hours: number analyzed (Participants) | 10 | 10
  Plateau ventilatory pressure at 32 hours | 23.2 [20.38 to 26.41] | 23.2 [20.44 to 26.55]
  Plateau ventilatory pressure at 36 hours: number analyzed (Participants) | 11 | 9
  Plateau ventilatory pressure at 36 hours | 23.4 [20.63 to 26.59] | 23.7 [20.55 to 27.29]
  Plateau ventilatory pressure at 42 hours: number analyzed (Participants) | 9 | 9
  Plateau ventilatory pressure at 42 hours | 24.8 [21.36 to 28.57] | 23.3 [20.18 to 26.82]
  Plateau ventilatory pressure at 48 hours: number analyzed (Participants) | 9 | 7
  Plateau ventilatory pressure at 48 hours | 23.6 [20.32 to 27.73] | 23.1 [20.10 to 27.18]
  Plateau ventilatory pressure at 48.5 hours: number analyzed (Participants) | 8 | 8
  Plateau ventilatory pressure at 48.5 hours | 23.1 [19.89 to 27.11] | 25.2 [22.01 to 29.38]
  Plateau ventilatory pressure at 49 hours: number analyzed (Participants) | 7 | 8
  Plateau ventilatory pressure at 49 hours | 22.8 [19.34 to 26.73] | 24.6 [21.44 to 28.66]
  Plateau ventilatory pressure at 50 hours: number analyzed (Participants) | 7 | 9
  Plateau ventilatory pressure at 50 hours | 22.3 [19.01 to 26.27] | 25.2 [21.93 to 29.33]
  Plateau ventilatory pressure at 52 hours: number analyzed (Participants) | 7 | 8
  Plateau ventilatory pressure at 52 hours | 23.9 [20.46 to 28.73] | 25.4 [22.00 to 29.64]
  Plateau ventilatory pressure at 54 hours: number analyzed (Participants) | 8 | 8
  Plateau ventilatory pressure at 54 hours | 23.1 [19.75 to 27.63] | 23.1 [20.06 to 26.94]
  Plateau ventilatory pressure at 56 hours: number analyzed (Participants) | 7 | 9
  Plateau ventilatory pressure at 56 hours | 23.2 [19.87 to 27.85] | 22.4 [19.50 to 25.86]
  Plateau ventilatory pressure at 60 hours: number analyzed (Participants) | 6 | 7
  Plateau ventilatory pressure at 60 hours | 22.5 [18.69 to 27.06] | 23.4 [20.18 to 26.99]
  Plateau ventilatory pressure at 66 hours: number analyzed (Participants) | 4 | 7
  Plateau ventilatory pressure at 66 hours | 24.5 [19.54 to 30.63] | 23.6 [20.10 to 27.69]
  Plateau ventilatory pressure at 72 hours: number analyzed (Participants) | 4 | 7
  Plateau ventilatory pressure at 72 hours | 21.7 [17.69 to 26.83] | 25.3 [21.52 to 29.52]
  Plateau ventilatory pressure at 168 hours: number analyzed (Participants) | 2 | 3
  Plateau ventilatory pressure at 168 hours | 15.1 [11.70 to 19.47] | 17.0 [14.62 to 20.30]
Statistical Analysis 1: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 0.5 hours; Test type: Superiority or Other; p = 0.2598, Bayesian repeated measures model; Ratio of Active/Placebo = 0.93, 95% CI 2-sided [0.752 to 1.215]
Statistical Analysis 2: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 1 hour; Test type: Superiority or Other; p = 0.3949, Bayesian repeated measures model; Ratio of Active/Placebo = 0.97, 95% CI 2-sided [0.783 to 1.273]
Statistical Analysis 3: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 2 hours; Test type: Superiority or Other; p = 0.4175, Bayesian repeated measures model; Ratio of Active/Placebo = 0.98, 95% CI 2-sided [0.791 to 1.294]
Statistical Analysis 4: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 4 hours; Test type: Superiority or Other; p = 0.4420, Bayesian repeated measures model; Ratio of Active/Placebo = 0.98, 95% CI 2-sided [0.806 to 1.292]
Statistical Analysis 5: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 6 hours; Test type: Superiority or Other; p = 0.4432, Bayesian repeated measures model; Ratio of Active/Placebo = 0.99, 95% CI 2-sided [0.811 to 1.262]
Statistical Analysis 6: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 8 hours; Test type: Superiority or Other; p = 0.4578, Bayesian repeated measures model; Ratio of Active/Placebo = 0.99, 95% CI 2-sided [0.818 to 1.229]
Statistical Analysis 7: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 12 hours; Test type: Superiority or Other; p = 0.3365, Bayesian repeated measures model; Ratio of Active/Placebo = 0.96, 95% CI 2-sided [0.790 to 1.167]
Statistical Analysis 8: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 18 hours; Test type: Superiority or Other; p = 0.3339, Bayesian repeated measures model; Ratio of Active/Placebo = 0.95, 95% CI 2-sided [0.770 to 1.163]
Statistical Analysis 9: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24 hours; Test type: Superiority or Other; p = 0.3608, Bayesian repeated measures model; Ratio of Active/Placebo = 0.96, 95% CI 2-sided [0.786 to 1.166]
Statistical Analysis 10: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24.5 hours; Test type: Superiority or Other; p = 0.3584, Bayesian repeated measures model; Ratio of Active/Placebo = 0.96, 95% CI 2-sided [0.788 to 1.168]
Statistical Analysis 11: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 25 hours; Test type: Superiority or Other; p = 0.1219, Bayesian repeated measures model; Ratio of Active/Placebo = 0.88, 95% CI 2-sided [0.725 to 1.073]
Statistical Analysis 12: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 26 hours; Test type: Superiority or Other; p = 0.4662, Bayesian repeated measures model; Ratio of Active/Placebo = 0.99, 95% CI 2-sided [0.814 to 1.210]
Statistical Analysis 13: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 28 hours; Test type: Superiority or Other; p = 0.5748, Bayesian repeated measures model; Ratio of Active/Placebo = 1.02, 95% CI 2-sided [0.828 to 1.247]
Statistical Analysis 14: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 30 hours; Test type: Superiority or Other; p = 0.4104, Bayesian repeated measures model; Ratio of Active/Placebo = 0.97, 95% CI 2-sided [0.786 to 1.204]
Statistical Analysis 15: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 32 hours; Test type: Superiority or Other; p = 0.5114, Bayesian repeated measures model; Ratio of Active/Placebo = 1.00, 95% CI 2-sided [0.817 to 1.246]
Statistical Analysis 16: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 36 hours; Test type: Superiority or Other; p = 0.4213, Bayesian repeated measures model; Ratio of Active/Placebo = 0.98, 95% CI 2-sided [0.783 to 1.200]
Statistical Analysis 17: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 42 hours; Test type: Superiority or Other; p = 0.2663, Bayesian repeated measures model; Ratio of Active/Placebo = 0.93, 95% CI 2-sided [0.731 to 1.132]
Statistical Analysis 18: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48 hours; Test type: Superiority or Other; p = 0.2373, Bayesian repeated measures model; Ratio of Active/Placebo = 0.91, 95% CI 2-sided [0.720 to 1.142]
Statistical Analysis 19: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48.5 hours; Test type: Superiority or Other; p = 0.2575, Bayesian repeated measures model; Ratio of Active/Placebo = 0.92, 95% CI 2-sided [0.721 to 1.149]
Statistical Analysis 20: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 49 hours; Test type: Superiority or Other; p = 0.2173, Bayesian repeated measures model; Ratio of Active/Placebo = 0.90, 95% CI 2-sided [0.708 to 1.127]
Statistical Analysis 21: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 50 hours; Test type: Superiority or Other; p = 0.2406, Bayesian repeated measures model; Ratio of Active/Placebo = 0.91, 95% CI 2-sided [0.717 to 1.143]
Statistical Analysis 22: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 52 hours; Test type: Superiority or Other; p = 0.2471, Bayesian repeated measures model; Ratio of Active/Placebo = 0.92, 95% CI 2-sided [0.721 to 1.151]
Statistical Analysis 23: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 54 hours; Test type: Superiority or Other; p = 0.2585, Bayesian repeated measures model; Ratio of Active/Placebo = 0.93, 95% CI 2-sided [0.727 to 1.157]
Statistical Analysis 24: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 56 hours; Test type: Superiority or Other; p = 0.3101, Bayesian repeated measures model; Ratio of Active/Placebo = 0.94, 95% CI 2-sided [0.737 to 1.170]
Statistical Analysis 25: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 60 hours; Test type: Superiority or Other; p = 0.2476, Bayesian repeated measures model; Ratio of Active/Placebo = 0.92, 95% CI 2-sided [0.727 to 1.160]
Statistical Analysis 26: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 66 hours; Test type: Superiority or Other; p = 0.3887, Bayesian repeated measures model; Ratio of Active/Placebo = 0.96, 95% CI 2-sided [0.767 to 1.222]
Statistical Analysis 27: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority; p = 0.2294, Bayesian repeated measures model; Ratio of Active/Placebo = 0.92, 95% CI 2-sided [0.749 to 1.146]
Statistical Analysis 28: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PEEP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 168 hours; Test type: Superiority or Other; p = 0.8522, Bayesian repeated measures model; Ratio of Active/Placebo = 1.09, 95% CI 2-sided [0.916 to 1.234]
Statistical Analysis 29: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 0.5 hours; Test type: Superiority or Other; p = 0.5885, Bayesian repeated measures model; Ratio of Active/Placebo = 1.02, 95% CI 2-sided [0.890 to 1.164]
Statistical Analysis 30: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 1 hour; Test type: Superiority or Other; p = 0.8558, Bayesian repeated measures model; Ratio of Active/Placebo = 1.07, 95% CI 2-sided [0.940 to 1.230]
Statistical Analysis 31: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 2 hour; Test type: Superiority or Other; p = 0.8374, Bayesian repeated measures model; Ratio of Active/Placebo = 1.07, 95% CI 2-sided [0.932 to 1.224]
Statistical Analysis 32: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 4 hours; Test type: Superiority or Other; p = 0.5886, Bayesian repeated measures model; Ratio of Active/Placebo = 1.01, 95% CI 2-sided [0.887 to 1.152]
Statistical Analysis 33: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 6 hours; Test type: Superiority or Other; p = 0.7532, Bayesian repeated measures model; Ratio of Active/Placebo = 1.05, 95% CI 2-sided [0.918 to 1.180]
Statistical Analysis 34: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 8 hours; Test type: Superiority or Other; p = 0.7108, Bayesian repeated measures model; Ratio of Active/Placebo = 1.04, 95% CI 2-sided [0.906 to 1.179]
Statistical Analysis 35: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 12 hours; Test type: Superiority or Other; p = 0.7445, Bayesian repeated measures model; Ratio of Active/Placebo = 1.04, 95% CI 2-sided [0.918 to 1.190]
Statistical Analysis 36: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 18 hours; Test type: Superiority or Other; p = 0.3759, Bayesian repeated measures model; Ratio of Active/Placebo = 0.98, 95% CI 2-sided [0.863 to 1.115]
Statistical Analysis 37: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24 hours; Test type: Superiority or Other; p = 0.3980, Bayesian repeated measures model; Ratio of Active/Placebo = 0.98, 95% CI 2-sided [0.859 to 1.118]
Statistical Analysis 38: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24.5 hours; Test type: Superiority or Other; p = 0.3231, Bayesian repeated measures model; Ratio of Active/Placebo = 0.97, 95% CI 2-sided [0.849 to 1.103]
Statistical Analysis 39: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 25 hours; Test type: Superiority or Other; p = 0.1245, Bayesian repeated measures model; Ratio of Active/Placebo = 0.93, 95% CI 2-sided [0.812 to 1.056]
Statistical Analysis 40: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 26 hours; Test type: Superiority or Other; p = 0.4631, Bayesian repeated measures model; Ratio of Active/Placebo = 0.99, 95% CI 2-sided [0.870 to 1.134]
Statistical Analysis 41: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 28 hours; Test type: Superiority or Other; p = 0.1026, Bayesian repeated measures model; Ratio of Active/Placebo = 0.92, 95% CI 2-sided [0.801 to 1.047]
Statistical Analysis 42: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 30 hours; Test type: Superiority or Other; p = 0.3152, Bayesian repeated measures model; Ratio of Active/Placebo = 0.97, 95% CI 2-sided [0.850 to 1.101]
Statistical Analysis 43: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 32 hours; Test type: Superiority or Other; p = 0.0762, Bayesian repeated measures model; Ratio of Active/Placebo = 0.91, 95% CI 2-sided [0.803 to 1.035]
Statistical Analysis 44: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 36 hours; Test type: Superiority or Other; p = 0.0274, Bayesian repeated measures model; Ratio of Active/Placebo = 0.88, 95% CI [0.763 to 1.003]
Statistical Analysis 45: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 42 hours; Test type: Superiority or Other; p = 0.3594, Bayesian repeated measures model; Ratio of Active/Placebo = 0.98, 95% CI 2-sided [0.853 to 1.112]
Statistical Analysis 46: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48 hours; Test type: Superiority or Other; p = 0.7027, Bayesian repeated measures model; Ratio of Active/Placebo = 1.04, 95% CI 2-sided [0.906 to 1.197]
Statistical Analysis 47: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48.5 hours; Test type: Superiority or Other; p = 0.8661, Bayesian repeated measures model; Ratio of Active/Placebo = 1.08, 95% CI 2-sided [0.941 to 1.246]
Statistical Analysis 48: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 49 hours; Test type: Superiority or Other; p = 0.8084, Bayesian repeated measures model; Ratio of Active/Placebo = 1.06, 95% CI 2-sided [0.924 to 1.228]
Statistical Analysis 49: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 50 hours; Test type: Superiority or Other; p = 0.9504, Bayesian repeated measures model; Ratio of Active/Placebo = 1.13, 95% CI 2-sided [0.976 to 1.300]
Statistical Analysis 50: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 52 hours; Test type: Superiority or Other; p = 0.5300, Bayesian repeated measures model; Ratio of Active/Placebo = 1.01, 95% CI 2-sided [0.871 to 1.164]
Statistical Analysis 51: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 54 hours; Test type: Superiority or Other; p = 0.8595, Bayesian repeated measures model; Ratio of Active/Placebo = 1.08, 95% CI 2-sided [0.942 to 1.243]
Statistical Analysis 52: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 56 hours; Test type: Superiority or Other; p = 0.8802, Bayesian repeated measures model; Ratio of Active/Placebo = 1.09, 95% CI 2-sided [0.943 to 1.261]
Statistical Analysis 53: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 60 hours; Test type: Superiority or Other; p = 0.9232, Bayesian repeated measures model; Ratio of Active/Placebo = 1.11, 95% CI 2-sided [0.958 to 1.278]
Statistical Analysis 54: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 66 hours; Test type: Superiority or Other; p = 0.7911, Bayesian repeated measures model; Ratio of Active/Placebo = 1.07, 95% CI 2-sided [0.902 to 1.256]
Statistical Analysis 55: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority or Other; p = 0.9946, Bayesian repeated measures model; Ratio of Active/Placebo = 1.28, 95% CI 2-sided [1.059 to 1.514]
Statistical Analysis 56: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Peak ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 168 hours; Test type: Superiority or Other; p = 0.9830, Bayesian repeated measures model; Ratio of Active/Placebo = 1.26, 95% CI 2-sided [1.019 to 1.444]
Statistical Analysis 57: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 0.5 hours; Test type: Superiority or Other; p = 0.8024, Bayesian repeated measures model; Ratio of Active/Placebo = 1.08, 95% CI 2-sided [0.910 to 1.261]
Statistical Analysis 58: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 1 hour; Test type: Superiority or Other; p = 0.4806, Bayesian repeated measures model; Ratio of Active/Placebo = 1.00, 95% CI 2-sided [0.843 to 1.166]
Statistical Analysis 59: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 2 hours; Test type: Superiority or Other; p = 0.6658, Bayesian repeated measures model; Ratio of Active/Placebo = 1.04, 95% CI 2-sided [0.869 to 1.223]
Statistical Analysis 60: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 4 hours; Test type: Superiority or Other; p = 0.6131, Bayesian repeated measures model; Ratio of Active/Placebo = 1.03, 95% CI 2-sided [0.856 to 1.212]
Statistical Analysis 61: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 6 hours; Test type: Superiority or Other; p = 0.5795, Bayesian repeated measures model; Ratio of Active/Placebo = 1.02, 95% CI 2-sided [0.856 to 1.197]
Statistical Analysis 62: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 8 hours; Test type: Superiority or Other; p = 0.0209, Bayesian repeated measures model; Ratio of Active/Placebo = 0.85, 95% CI 2-sided [0.716 to 0.993]
Statistical Analysis 63: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 12 hours; Test type: Superiority or Other; p = 0.4823, Mixed Models Analysis; Ratio of Active/Placebo = 1.00, 95% CI 2-sided [0.830 to 1.187]
Statistical Analysis 64: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 18 hours; Test type: Superiority or Other; p = 0.0406, Bayesian repeated measures model; 0.0406 = 0.85, 95% CI 2-sided [0.703 to 1.021]
Statistical Analysis 65: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24 hours; Test type: Superiority or Other; p = 0.5186, Bayesian repeated measures model; Ratio of Active/Placebo = 1.00, 95% CI 2-sided [0.844 to 1.169]
Statistical Analysis 66: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24.5 hours; Test type: Superiority or Other; p = 0.3870, Bayesian repeated measures model; Ratio of Active/Placebo = 0.98, 95% CI 2-sided [0.824 to 1.132]
Statistical Analysis 67: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 25 hours; Test type: Superiority or Other; p = 0.1281, Bayesian repeated measures model; Ratio of Active/Placebo = 0.91, 95% CI 2-sided [0.770 to 1.065]
Statistical Analysis 68: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 26 hours; Test type: Superiority or Other; p = 0.4754, Bayesian repeated measures model; Ratio of Active/Placebo = 0.99, 95% CI 2-sided [0.837 to 1.181]
Statistical Analysis 69: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 28 hours; Test type: Superiority or Other; p = 0.5627, Bayesian repeated measures model; Ratio of Active/Placebo = 1.01, 95% CI 2-sided [0.856 to 1.217]
Statistical Analysis 70: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 30 hours; Test type: Superiority or Other; p = 0.5552, Bayesian repeated measures model; Ratio of Active/Placebo = 1.01, 95% CI 2-sided [0.848 to 1.220]
Statistical Analysis 71: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 32 hours; Test type: Superiority or Other; p = 0.5030, Bayesian repeated measures model; Ratio of Active/Placebo = 1.00, 95% CI 2-sided [0.843 to 1.201]
Statistical Analysis 72: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 36 hours; Test type: Superiority or Other; p = 0.5558, Bayesian repeated measures model; Ratio of Active/Placebo = 1.01, 95% CI 2-sided [0.840 to 1.218]
Statistical Analysis 73: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 42 hours; Test type: Superiority or Other; p = 0.2709, Bayesian repeated measures model; Ratio of Active/Placebo = 0.94, 95% CI 2-sided [0.769 to 1.135]
Statistical Analysis 74: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48 hours; Test type: Superiority or Other; p = 0.4143, Bayesian repeated measures model; Ratio of Active/Placebo = 0.98, 95% CI 2-sided [0.795 to 1.208]
Statistical Analysis 75: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48.5 hours; Test type: Superiority or Other; p = 0.7886, Bayesian repeated measures model; Ratio of Active/Placebo = 1.09, 95% CI 2-sided [0.891 to 1.348]
Statistical Analysis 76: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 49 hours; Test type: Superiority or Other; p = 0.7607, Bayesian repeated measures model; Ratio of Active/Placebo = 1.08, 95% CI 2-sided [0.885 to 1.353]
Statistical Analysis 77: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 50 hours; Test type: Superiority or Other; p = 0.8677, Bayesian repeated measures model; Ratio of Active/Placebo = 1.13, 95% CI 2-sided [0.922 to 1.400]
Statistical Analysis 78: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 52 hours; Test type: Superiority or Other; p = 0.7012, Bayesian repeated measures model; Ratio of Active/Placebo = 1.06, 95% CI 2-sided [0.847 to 1.302]
Statistical Analysis 79: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 54 hours; Test type: Superiority or Other; p = 0.5156, Bayesian repeated measures model; Ratio of Active/Placebo = 1.00, 95% CI 2-sided [0.805 to 1.230]
Statistical Analysis 80: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 56 hours; Test type: Superiority or Other; p = 0.3524, Bayesian repeated measures model; Ratio of Active/Placebo = 0.96, 95% CI 2-sided [0.783 to 1.178]
Statistical Analysis 81: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 60 hours; Test type: Superiority or Other; p = 0.6380, Bayesian repeated measures model; Ratio of Active/Placebo = 1.04, 95% CI 2-sided [0.845 to 1.292]
Statistical Analysis 82: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 66 hours; Test type: Superiority or Other; p = 0.4003, Bayesian repeated measures model; Ratio of Active/Placebo = 0.96, 95% CI 2-sided [0.743 to 1.241]
Statistical Analysis 83: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority or Other; p = 0.8817, Bayesian repeated measures model; Ratio of Active/Placebo = 1.16, 95% CI 2-sided [0.907 to 1.502]
Statistical Analysis 84: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Plateau ventilatory pressure, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 168 hours; Test type: Superiority or Other; p = 0.8145, Bayesian repeated measures model; Ratio of Active/Placebo = 1.14, 95% CI 2-sided [0.804 to 1.505]

25. Secondary Outcome: Measure of Oxygenation Including Fraction of Inspired Oxygen/ Partial Pressure of Oxygen in Arterial Blood (PaO2/FiO2) Ratio Via Pulse Oximetry Upto Day 7 (Part B)
Description: Measure of oxygenation included PaO2/FiO2 ratio defined as the ratio of arterial oxygen partial pressure to fractional inspired oxygen by pulse oximeter a device that measured the oxygen saturation of arterial blood in a participant by utilizing a sensor attached typically to a finger, toe, or ear to determine the percentage of oxyhemoglobin in blood pulsating through a network of capillaries.
  Assessments were performed at 0.5, 1, 2, 4, 6, 8, 12, 18, 24, 24.5, 25, 26, 28, 30, 32, 36, 42, 48, 48.5, 49, 50, 52, 54, 56, 60, 66, 72 and 168 hours upto Day 7. Data has been presented for median along with the 95% credible interval.
Time Frame: as for outcome 24
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Median (95% Confidence Interval); unit: Ratio
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
Ratio
  PaO2/FiO2 at 0.5 hours: number analyzed (Participants) | 18 | 17
  PaO2/FiO2 at 0.5 hours | 166.2 [139.71 to 201.29] | 173.7 [143.97 to 206.37]
  PaO2/FiO2 at 1 hour: number analyzed (Participants) | 17 | 16
  PaO2/FiO2 at 1 hour | 178.1 [149.67 to 215.96] | 160.2 [132.71 to 190.93]
  PaO2/FiO2 at 2 hours: number analyzed (Participants) | 20 | 18
  PaO2/FiO2 at 2 hours | 181.5 [153.14 to 216.76] | 162.3 [137.17 to 192.34]
  PaO2/FiO2 at 4 hours: number analyzed (Participants) | 19 | 17
  PaO2/FiO2 at 4 hours | 182.8 [153.78 to 218.35] | 155.1 [130.45 to 183.88]
  PaO2/FiO2 at 6 hours: number analyzed (Participants) | 20 | 18
  PaO2/FiO2 at 6 hours | 173.2 [146.00 to 205.32] | 156.7 [130.95 to 186.82]
  PaO2/FiO2 at 8 hours: number analyzed (Participants) | 19 | 18
  PaO2/FiO2 at 8 hours | 160.9 [135.62 to 191.40] | 170.6 [143.85 to 203.91]
  PaO2/FiO2 at 12 hours: number analyzed (Participants) | 18 | 17
  PaO2/FiO2 at 12 hours | 173.7 [144.53 to 208.14] | 179.6 [149.68 to 214.58]
  PaO2/FiO2 at 18 hours: number analyzed (Participants) | 19 | 18
  PaO2/FiO2 at 18 hours | 180.5 [151.11 to 214.80] | 176.8 [147.25 to 212.12]
  PaO2/FiO2 at 24 hours: number analyzed (Participants) | 17 | 19
  PaO2/FiO2 at 24 hours | 183.5 [153.03 to 219.67] | 167.3 [141.36 to 199.09]
  PaO2/FiO2 at 24.5 hours: number analyzed (Participants) | 18 | 17
  PaO2/FiO2 at 24.5 hours | 189.3 [158.67 to 226.84] | 175.8 [147.94 to 209.31]
  PaO2/FiO2 at 25 hours: number analyzed (Participants) | 17 | 18
  PaO2/FiO2 at 25 hours | 179.6 [150.61 to 215.78] | 167.1 [139.64 to 198.81]
  PaO2/FiO2 at 26 hours: number analyzed (Participants) | 18 | 18
  PaO2/FiO2 at 26 hours | 182.9 [153.39 to 219.07] | 183.2 [153.67 to 217.68]
  PaO2/FiO2 at 28 hours: number analyzed (Participants) | 18 | 17
  PaO2/FiO2 at 28 hours | 191.1 [159.67 to 229.27] | 167.9 [140.69 to 200.46]
  PaO2/FiO2 at 30 hours: number analyzed (Participants) | 17 | 17
  PaO2/FiO2 at 30 hours | 169.5 [140.90 to 205.06] | 169.3 [139.80 to 204.89]
  PaO2/FiO2 at 32 hours: number analyzed (Participants) | 17 | 18
  PaO2/FiO2 at 32 hours | 174.2 [143.12 to 210.61] | 155.3 [128.84 to 186.13]
  PaO2/FiO2 at 36 hours: number analyzed (Participants) | 17 | 19
  PaO2/FiO2 at 36 hours | 200.5 [164.55 to 240.83] | 159.5 [132.90 to 191.36]
  PaO2/FiO2 at 42 hours: number analyzed (Participants) | 17 | 18
  PaO2/FiO2 at 42 hours | 172.7 [142.65 to 207.00] | 171.0 [143.95 to 203.01]
  PaO2/FiO2 at 48 hours: number analyzed (Participants) | 14 | 18
  PaO2/FiO2 at 48 hours | 169.9 [139.20 to 206.04] | 178.2 [148.82 to 214.14]
  PaO2/FiO2 at 48.5 hours: number analyzed (Participants) | 14 | 18
  PaO2/FiO2 at 48.5 hours | 195.8 [159.95 to 237.96] | 175.5 [146.24 to 211.20]
  PaO2/FiO2 at 49 hours: number analyzed (Participants) | 13 | 17
  PaO2/FiO2 at 49 hours | 166.5 [135.67 to 203.47] | 175.1 [144.85 to 211.61]
  PaO2/FiO2 at 50 hours: number analyzed (Participants) | 14 | 16
  PaO2/FiO2 at 50 hours | 168.3 [138.07 to 205.14] | 167.5 [137.42 to 202.44]
  PaO2/FiO2 at 52 hours: number analyzed (Participants) | 13 | 18
  PaO2/FiO2 at 52 hours | 183.9 [149.96 to 227.12] | 168.4 [141.57 to 202.76]
  PaO2/FiO2 at 54 hours: number analyzed (Participants) | 14 | 17
  PaO2/FiO2 at 54 hours | 191.6 [156.36 to 235.76] | 172.1 [144.47 to 204.97]
  PaO2/FiO2 at 56 hours: number analyzed (Participants) | 13 | 17
  PaO2/FiO2 at 56 hours | 181.6 [148.45 to 224.06] | 173.9 [146.20 to 206.22]
  PaO2/FiO2 at 60 hours: number analyzed (Participants) | 14 | 18
  PaO2/FiO2 at 60 hours | 170.8 [139.25 to 210.58] | 162.4 [135.34 to 192.99]
  PaO2/FiO2 at 66 hours: number analyzed (Participants) | 15 | 17
  PaO2/FiO2 at 66 hours | 154.6 [126.25 to 189.63] | 162.6 [133.81 to 195.44]
  PaO2/FiO2 at 72 hours: number analyzed (Participants) | 11 | 18
  PaO2/FiO2 at 72 hours | 150.4 [119.68 to 188.02] | 153.3 [128.23 to 183.15]
  PaO2/FiO2 at 168 hours: number analyzed (Participants) | 8 | 10
  PaO2/FiO2 at 168 hours | 198.9 [163.04 to 266.41] | 168.9 [143.77 to 196.40]
Statistical Analysis 1: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 0.5 hours; Test type: Superiority or Other; p = 0.6468, Bayesian repeated measures model; Ratio of Active/Placebo = 1.05, 95% CI 2-sided [0.765 to 1.321]
Statistical Analysis 2: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 1 hour; Test type: Superiority or Other; p = 0.1965, Bayesian repeated measures model; Ratio of Active/Placebo = 0.90, 95% CI 2-sided [0.658 to 1.136]
Statistical Analysis 3: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 2 hours; Test type: Superiority or Other; p = 0.1681, Bayesian repeated measures model; Ratio of Active/Placebo = 0.90, 95% CI 2-sided [0.694 to 1.129]
Statistical Analysis 4: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 4 hours; Test type: Superiority or Other; p = 0.0877, Bayesian repeated measures model; Ratio of Active/Placebo = 0.85, 95% CI 2-sided [0.669 to 1.075]
Statistical Analysis 5: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 6 hours; Test type: Superiority or Other; p = 0.2011, Bayesian repeated measures model; Ratio of Active/Placebo = 0.90, 95% CI 2-sided [0.715 to 1.159]
Statistical Analysis 6: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 8 hours; Test type: Superiority or Other; p = 0.6855, Bayesian repeated measures model; Ratio of Active/Placebo = 1.06, 95% CI 2-sided [0.842 to 1.345]
Statistical Analysis 7: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 12 hours; Test type: Superiority or Other; p = 0.6093, Bayesian repeated measures model; Ratio of Active/Placebo = 1.04, 95% CI 2-sided [0.800 to 1.325]
Statistical Analysis 8: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 18 hours; Test type: Superiority or Other; p = 0.4350, Bayesian repeated measures model; Ratio of Active/Placebo = 0.98, 95% CI 2-sided [0.765 to 1.253]
Statistical Analysis 9: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24 hours; Test type: Superiority or Other; p = 0.2232, Bayesian repeated measures model; Ratio of Active/Placebo = 0.91, 95% CI 2-sided [0.722 to 1.195]
Statistical Analysis 10: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24.5 hours; Test type: Superiority or Other; p = 0.2716, Bayesian repeated measures model; Ratio of Active/Placebo = 0.93, 95% CI 2-sided [0.733 to 1.200]
Statistical Analysis 11: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 25 hours; Test type: Superiority or Other; p = 0.2866, Bayesian repeated measures model; Ratio of Active/Placebo = 0.93, 95% CI 2-sided [0.726 to 1.190]
Statistical Analysis 12: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 26 hours; Test type: Superiority or Other; p = 0.5033, Bayesian repeated measures model; Ratio of Active/Placebo = 1.00, 95% CI 2-sided [0.780 to 1.270]
Statistical Analysis 13: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 28 hours; Test type: Superiority or Other; p = 0.1493, Bayesian repeated measures model; Ratio of Active/Placebo = 0.88, 95% CI 2-sided [0.684 to 1.120]
Statistical Analysis 14: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 30 hours; Test type: Superiority or Other; p = 0.4947, Bayesian repeated measures model; Ratio of Active/Placebo = 1.00, 95% CI 2-sided [0.759 to 1.301]
Statistical Analysis 15: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 32 hours; Test type: Superiority or Other; p = 0.1951, Bayesian repeated measures model; Ratio of Active/Placebo = 0.89, 95% CI 2-sided [0.678 to 1.161]
Statistical Analysis 16: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 36 hours; Test type: Superiority or Other; p = 0.0512, Bayesian repeated measures model; Ratio of Active/Placebo = 0.80, 95% CI 2-sided [0.612 to 1.050]
Statistical Analysis 17: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 42 hours; Test type: Superiority or Other; p = 0.4700, Bayesian repeated measures model; Ratio of Active/Placebo = 0.99, 95% CI 2-sided [0.775 to 1.279]
Statistical Analysis 18: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48 hours; Test type: Superiority or Other; p = 0.6340, Bayesian repeated measures model; Ratio of Active/Placebo = 1.05, 95% CI 2-sided [0.811 to 1.368]
Statistical Analysis 19: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48.5 hours; Test type: Superiority or Other; p = 0.2129, Bayesian repeated measures model; Ratio of Active/Placebo = 0.90, 95% CI 2-sided [0.689 to 1.183]
Statistical Analysis 20: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 49 hours; Test type: Superiority or Other; p = 0.6418, Bayesian repeated measures model; Ratio of Active/Placebo = 1.05, 95% CI 2-sided [0.798 to 1.411]
Statistical Analysis 21: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 50 hours; Test type: Superiority or Other; p = 0.4797, Ratio of Active/Placebo; Ratio of Active/Placebo = 0.99, 95% CI 2-sided [0.754 to 1.315]
Statistical Analysis 22: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 52 hours; Test type: Superiority or Other; p = 0.2659, Bayesian repeated measures model; Ratio of Active/Placebo = 0.92, 95% CI 2-sided [0.703 to 1.199]
Statistical Analysis 23: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 54 hours; Test type: Superiority or Other; p = 0.2102, Bayesian repeated measures model; Ratio of Active/Placebo = 0.90, 95% CI 2-sided [0.687 to 1.159]
Statistical Analysis 24: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 56 hours; Test type: Superiority or Other; p = 0.3623, Bayesian repeated measures model; Ratio of Active/Placebo = 0.96, 95% CI 2-sided [0.740 to 1.240]
Statistical Analysis 25: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 60 hours; Test type: Superiority or Other; p = 0.3499, Bayesian repeated measures model; Ratio of Active/Placebo = 0.95, 95% CI 2-sided [0.730 to 1.225]
Statistical Analysis 26: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 66 hours; Test type: Superiority or Other; p = 0.6494, Bayesian repeated measures model; Ratio of Active/Placebo = 1.05, 95% CI 2-sided [0.787 to 1.377]
Statistical Analysis 27: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority or Other; p = 0.5567, Bayesian repeated measures model; Ratio of Active/Placebo = 1.02, 95% CI 2-sided [0.766 to 1.358]
Statistical Analysis 28: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); PaO2/FiO2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 168 hours; Test type: Superiority or Other; p = 0.1095, Bayesian repeated measures model; Ratio of Active/Placebo = 0.85, 95% CI 2-sided [0.615 to 1.073]

26. Secondary Outcome: Measure of Oxygenation Index Upto Day 7 (Part B)
Description: Oxygenation index was defined as calculation used in intensive care medicine to measure the fraction of inspired oxygen (FiO2) and its usage within the body and was computed using the equation Oxygenation Index= FiO2 x Mean Airway Pressure/Pao2. Assessments were performed at 0.5, 1, 2, 4, 6, 8, 12, 18, 24, 24.5, 25, 26, 28, 30, 32, 36, 42, 48, 48.5, 49, 50, 52, 54, 56, 60, 66, 72 and 168 hours upto Day 7. Data has been presented for median along with the 95% credible interval.
Time Frame: as for outcome 24
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Median (95% Confidence Interval); unit: Percentage
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
Percentage
  Oxygenation index at 0.5 hours: number analyzed (Participants) | 16 | 15
  Oxygenation index at 0.5 hours | 10.0 [7.26 to 13.17] | 10.6 [7.71 to 14.79]
  Oxygenation index at 1 hour: number analyzed (Participants) | 15 | 12
  Oxygenation index at 1 hour | 9.0 [6.60 to 11.82] | 12.2 [8.95 to 16.99]
  Oxygenation index at 2 hours: number analyzed (Participants) | 16 | 13
  Oxygenation index at 2 hours | 9.9 [7.35 to 12.96] | 11.0 [7.95 to 15.15]
  Oxygenation index at 4 hours: number analyzed (Participants) | 15 | 12
  Oxygenation index at 4 hours | 9.3 [7.01 to 12.43] | 11.6 [8.27 to 16.97]
  Oxygenation index at 6 hours: number analyzed (Participants) | 17 | 12
  Oxygenation index at 6 hours | 10.2 [7.65 to 13.46] | 12.3 [8.65 to 18.07]
  Oxygenation index at 8 hours: number analyzed (Participants) | 17 | 12
  Oxygenation index at 8 hours | 10.4 [7.76 to 13.89] | 12.4 [8.86 to 17.36]
  Oxygenation index at 12 hours: number analyzed (Participants) | 16 | 11
  Oxygenation index at 12 hours | 9.3 [6.88 to 12.61] | 11.0 [7.50 to 16.24]
  Oxygenation index at 18 hours: number analyzed (Participants) | 16 | 11
  Oxygenation index at 18 hours | 8.7 [6.44 to 11.52] | 10.8 [7.54 to 16.17]
  Oxygenation index at 24 hours: number analyzed (Participants) | 16 | 14
  Oxygenation index at 24 hours | 10.6 [8.02 to 14.05] | 10.6 [8.22 to 14.39]
  Oxygenation index at 24.5 hours: number analyzed (Participants) | 18 | 13
  Oxygenation index at 24.5 hours | 9.0 [6.79 to 11.90] | 9.6 [7.52 to 13.14]
  Oxygenation index at 25 hours: number analyzed (Participants) | 16 | 13
  Oxygenation index at 25 hours | 8.9 [6.74 to 11.93] | 10.5 [8.26 to 14.59]
  Oxygenation index at 26 hours: number analyzed (Participants) | 16 | 13
  Oxygenation index at 26 hours | 9.2 [6.92 to 12.16] | 8.3 [6.46 to 11.75]
  Oxygenation index at 28 hours: number analyzed (Participants) | 17 | 12
  Oxygenation index at 28 hours | 9.0 [6.86 to 12.01] | 9.4 [6.95 to 13.27]
  Oxygenation index at 30 hours: number analyzed (Participants) | 15 | 14
  Oxygenation index at 30 hours | 9.8 [7.42 to 13.33] | 9.6 [7.23 to 13.14]
  Oxygenation index at 32 hours: number analyzed (Participants) | 15 | 14
  Oxygenation index at 32 hours | 9.7 [7.21 to 13.16] | 10.4 [7.61 to 14.11]
  Oxygenation index at 36 hours: number analyzed (Participants) | 16 | 13
  Oxygenation index at 36 hours | 8.7 [6.31 to 11.81] | 10.1 [7.29 to 13.79]
  Oxygenation index at 42 hours: number analyzed (Participants) | 16 | 13
  Oxygenation index at 42 hours | 9.4 [6.98 to 12.70] | 10.2 [7.13 to 14.75]
  Oxygenation index at 48 hours: number analyzed (Participants) | 13 | 13
  Oxygenation index at 48 hours | 10.2 [7.58 to 14.29] | 8.8 [6.49 to 13.06]
  Oxygenation index at 48.5 hours: number analyzed (Participants) | 13 | 12
  Oxygenation index at 48.5 hours | 9.2 [6.78 to 12.79] | 8.4 [6.25 to 12.37]
  Oxygenation index at 49 hours: number analyzed (Participants) | 12 | 12
  Oxygenation index at 49 hours | 10.8 [7.90 to 15.04] | 8.9 [6.67 to 12.91]
  Oxygenation index at 50 hours: number analyzed (Participants) | 12 | 12
  Oxygenation index at 50 hours | 10.4 [7.63 to 14.64] | 9.2 [6.84 to 12.96]
  Oxygenation index at 52 hours: number analyzed (Participants) | 12 | 12
  Oxygenation index at 52 hours | 9.8 [7.07 to 13.78] | 9.4 [6.68 to 13.10]
  Oxygenation index at 54 hours: number analyzed (Participants) | 13 | 10
  Oxygenation index at 54 hours | 9.4 [6.83 to 12.99] | 9.7 [6.32 to 13.92]
  Oxygenation index at 56 hours: number analyzed (Participants) | 12 | 10
  Oxygenation index at 56 hours | 9.3 [6.86 to 12.97] | 8.5 [5.75 to 12.35]
  Oxygenation index at 60 hours: number analyzed (Participants) | 12 | 11
  Oxygenation index at 60 hours | 8.9 [6.33 to 12.53] | 9.9 [6.92 to 14.34]
  Oxygenation index at 66 hours: number analyzed (Participants) | 11 | 10
  Oxygenation index at 66 hours | 10.5 [7.27 to 14.66] | 8.2 [5.59 to 12.88]
  Oxygenation index at 72 hours: number analyzed (Participants) | 7 | 11
  Oxygenation index at 72 hours | 10.5 [6.62 to 16.36] | 9.7 [6.63 to 13.41]
  Oxygenation index at 168 hours: number analyzed (Participants) | 4 | 4
  Oxygenation index at 168 hours | 5.8 [4.31 to 9.67] | 6.4 [4.38 to 9.34]
Statistical Analysis 1: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 0.5 hours; Test type: Superiority or Other; p = 0.6098, Bayesian repeated measures model; Ratio of Active/Placebo = 1.06, 95% CI 2-sided [0.721 to 1.644]
Statistical Analysis 2: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 1 hour; Test type: Superiority or Other; p = 0.9441, Bayesian repeated measures model; Ratio of Active/Placebo = 1.35, 95% CI 2-sided [0.931 to 2.068]
Statistical Analysis 3: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 2 hours; Test type: Superiority or Other; p = 0.7173, Bayesian repeated measures model; Ratio of Active/Placebo = 1.12, 95% CI 2-sided [0.749 to 1.621]
Statistical Analysis 4: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 4 hours; Test type: Superiority or Other; p = 0.8292, Bayesian repeated measures model; Ratio of Active/Placebo = 1.26, 95% CI 2-sided [0.810 to 1.949]
Statistical Analysis 5: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 6 hours; Test type: Superiority or Other; p = 0.8008, Bayesian repeated measures model; Ratio of Active/Placebo = 1.23, 95% CI 2-sided [0.775 to 1.832]
Statistical Analysis 6: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 8 hours; Test type: Superiority or Other; p = 0.7905, Bayesian repeated measures model; Ratio of Active/Placebo = 1.20, 95% CI 2-sided [0.776 to 1.799]
Statistical Analysis 7: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 12 hours; Test type: Superiority or Other; p = 0.7566, Bayesian repeated measures model; Ratio of Active/Placebo = 1.17, 95% CI 2-sided [0.737 to 1.958]
Statistical Analysis 8: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 18 hours; Test type: Superiority or Other; p = 0.8349, Bayesian repeated measures model; Ratio of Active/Placebo = 1.25, 95% CI 2-sided [0.812 to 2.050]
Statistical Analysis 9: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24 hours; Test type: Superiority or Other; p = 0.4739, Bayesian repeated measures model; Ratio of Active/Placebo = 0.99, 95% CI 2-sided [0.713 to 1.527]
Statistical Analysis 10: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24.5 hours; Test type: Superiority or Other; p = 0.6291, Bayesian repeated measures model; Ratio of Active/Placebo = 1.06, 95% CI 2-sided [0.763 to 1.647]
Statistical Analysis 11: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 25 hours; Test type: Superiority or Other; p = 0.8032, Bayesian repeated measures model; Ratio of Active/Placebo = 1.18, 95% CI 2-sided [0.830 to 1.814]
Statistical Analysis 12: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 26 hours; Test type: Superiority or Other; p = 0.3250, Bayesian repeated measures model; Ratio of Active/Placebo = 0.91, 95% CI 2-sided [0.626 to 1.416]
Statistical Analysis 13: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 28 hours; Test type: Superiority or Other; p = 0.5828, Bayesian repeated measures model; Ratio of Active/Placebo = 1.05, 95% CI 2-sided [0.687 to 1.630]
Statistical Analysis 14: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 30 hours; Test type: Superiority or Other; p = 0.4546, Bayesian repeated measures model; Ratio of Active/Placebo = 0.98, 95% CI 2-sided [0.661 to 1.512]
Statistical Analysis 15: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 32 hours; Test type: Superiority or Other; p = 0.6158, Bayesian repeated measures model; Ratio of Active/Placebo = 1.06, 95% CI 2-sided [0.719 to 1.639]
Statistical Analysis 16: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 36 hours; Test type: Superiority or Other; p = 0.7748, Bayesian repeated measures model; Ratio of Active/Placebo = 1.17, 95% CI 2-sided [0.752 to 1.770]
Statistical Analysis 17: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 42 hours; Test type: Superiority or Other; p = 0.6565, Bayesian repeated measures model; Ratio of Active/Placebo = 1.09, 95% CI 2-sided [0.686 to 1.714]
Statistical Analysis 18: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48 hours; Test type: Superiority or Other; p = 0.2773, Bayesian repeated measures model; Ratio of Active/Placebo = 0.87, 95% CI 2-sided [0.566 to 1.380]
Statistical Analysis 19: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48.5 hours; Test type: Superiority or Other; p = 0.3606, Bayesian repeated measures model; Ratio of Active/Placebo = 0.92, 95% CI 2-sided [0.610 to 1.467]
Statistical Analysis 20: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 49 hours; Test type: Superiority or Other; p = 0.2211, Bayesian repeated measures model; Ratio of Active/Placebo = 0.83, 95% CI 2-sided [0.555 to 1.317]
Statistical Analysis 21: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 50 hours; Test type: Superiority or Other; p = 0.2860, Bayesian repeated measures model; Ratio of Active/Placebo = 0.88, 95% CI 2-sided [0.587 to 1.348]
Statistical Analysis 22: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 52 hours; Test type: Superiority or Other; p = 0.4079, Bayesian repeated measures model; Ratio of Active/Placebo = 0.94, 95% CI 2-sided [0.609 to 1.510]
Statistical Analysis 23: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 54 hours; Test type: Superiority or Other; p = 0.5284, Bayesian repeated measures model; Ratio of Active/Placebo = 1.02, 95% CI 2-sided [0.614 to 1.663]
Statistical Analysis 24: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 56 hours; Test type: Superiority or Other; p = 0.3586, Bayesian repeated measures model; Ratio of Active/Placebo = 0.90, 95% CI 2-sided [0.568 to 1.458]
Statistical Analysis 25: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 60 hours; Test type: Superiority or Other; p = 0.6768, Bayesian repeated measures model; Ratio of Active/Placebo = 1.13, 95% CI 2-sided [0.672 to 1.853]
Statistical Analysis 26: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 66 hours; Test type: Superiority or Other; p = 0.1574, Bayesian repeated measures model; Ratio of Active/Placebo = 0.77, 95% CI 2-sided [0.488 to 1.390]
Statistical Analysis 27: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority or Other; p = 0.3900, Bayesian repeated measures model; Ratio of Active/Placebo = 0.92, 95% CI 2-sided [0.521 to 1.584]
Statistical Analysis 28: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Oxygenation index, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 168 hours; Test type: Superiority or Other; p = 0.5915, Bayesian repeated measures model; Ratio of Active/Placebo = 1.05, 95% CI 2-sided [0.748 to 1.516]

27. Secondary Outcome: Number of Participants With Acute Kidney Injury as Defined by Day 1 to Day 3 Change in Risk, Injury, Failure, Loss of Kidney Function, and End-stage Kidney Disease (RIFLE) Criteria Upto Day 3 (Part B)
Description: The RIFLE score is made up of the glomerular filtration rate criteria (GFRC) and urine output criteria (UOC) and is defined as Risk (Serum Creatinine x 1.5 or GFR decrease > 25%-GFRC and < 0.5 milliliter/kilograms/hour [ml/kg/hour] x 6 hours-UOC), Injury (Serum Creatinine x 2 or GFR decrease > 50%-GFRC and < 0.5 ml/kg/hour x 12 hours), Failure (Serum Creatinine x 3, or GFR decrease > 75% [F=Failure] or Serum Creatinine >=4 milligrams/deciliter [mg/dl] with an acute rise > 0.5 mg/dl [Fc=Failure acute on chronic] and < 0.3 ml/kg/hour x 24 hours, or anuria x 12 hours [Fo=Failure oligouria]). Due to the duration of this study it was not possible to be calculate the designated RIFLE class Loss and RIFLE class End-stage kidney disease. Data has been presented for rifle score total, rifle score GFR and rifle score urine. Abbreviations NAKI= No acute kidney injury, R=risk, I=injury, MISS= Unable to derive score.
Time Frame: Upto Day 3
Population: The All Subjects - Part B Population.
Measure: Number; unit: Participants
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
Participants
  Rifle score total, MISS | 15 | 14
  Rifle score total, NAKI to NAKI | 3 | 1
  Rifle score total, NAKI to R | 1 | 0
  Rifle score total, R to NAKI | 1 | 1
  Rifle score total, I to NAKI | 0 | 1
  Rifle score total, I to I | 0 | 1
  Rifle score total, Fo to I | 0 | 1
  Rifle score GFR, MISS | 15 | 14
  Rifle score GFR, NAKI to NAKI | 5 | 2
  Rifle score GFR, R to I | 0 | 1
  Rifle score GFR, I to NAKI | 0 | 1
  Rifle score GFR, I to I | 0 | 1
  Rifle score urine, NAKI to NAKI | 10 | 11
  Rifle score urine, NAKI to Fo | 0 | 1
  Rifle score urine, NAKI to R | 2 | 0
  Rifle score urine, NAKI to I | 2 | 0
  Rifle score urine, R to NAKI | 1 | 2
  Rifle score urine, I to NAKI | 3 | 2
  Rifle score urine, I to R | 0 | 1
  Rifle score urine, Fo to NAKI | 1 | 0
  Rifle score urine, Fo to R | 0 | 1
  Rifle score urine, Fo to Fo | 1 | 1

28. Secondary Outcome: Evaluation of Sequential Organ Failure Assessment (SOFA) Score on Day 4 and Day 7 (Part B)
Description: The SOFA score is a mortality prediction score that is based on the degree of dysfunction of 6 organ systems (respiratory, nervous, cardiovascular, liver, coagulation, and kidneys). The score ranges from 0-24. 0 (normal) to 4 (high degree of dysfunction) is given for each organ system, with a higher score indicating greater severity. A score of 0-6 is associated with a mortality rate of less than 10% while a score between 16 and 24 is associated with a greater than 90% mortality rate.
Time Frame: Day 4 and Day 7
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (95% Confidence Interval); unit: Score on scale
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
Score on scale
  Total SOFA Score at Day 4: number analyzed (Participants) | 10 | 16
  Total SOFA Score at Day 4 | 7.4 [5.2 to 9.6] | 8.0 [6.3 to 9.7]
  Total SOFA Score at Day 7: number analyzed (Participants) | 7 | 6
  Total SOFA Score at Day 7 | 5.4 [2.7 to 8.2] | 6.8 [4.1 to 9.5]

29. Secondary Outcome: Biomarker Analysis for Serum Inflammatory Biomarkers, Markers of Neutrophil Activation, Markers of Lung Epithelial Cell Injury, Renin Levels and Aldosterone Levels Upto Day 5 (Part B)
Description: Serum inflammatory biomarkers included CXCL-8 [IL-8], IL-6, markers of neutrophil activation included (e.g. myeloperoxidase [MPO]), markers of lung epithelial cell injury included receptor for advanced glycation end-products [RAGE], Angiopoietin 2, along with rennin, aldosterone levels. Blood samples for biomarker analyses were collected 12 hours, 24 hours, 48 hours, 72 hours and 120 hours upto Day 5. Data has been presented for median along with the 95% credible interval.
Time Frame: 12 hours, 24 hours, 48 hours, 72 hours and 120 hours upto Day 5
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Median (95% Confidence Interval); unit: picograms per milliliter
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
picograms per milliliter
  CXCL-8 (IL-8) at 12 hours: number analyzed (Participants) | 14 | 18
  CXCL-8 (IL-8) at 12 hours | 18.7 [12.21 to 28.51] | 16.6 [11.73 to 23.39]
  CXCL-8 (IL-8) at 24 hours: number analyzed (Participants) | 13 | 17
  CXCL-8 (IL-8) at 24 hours | 17.5 [11.52 to 26.66] | 16.8 [11.94 to 23.57]
  CXCL-8 (IL-8) at 48 hours: number analyzed (Participants) | 11 | 15
  CXCL-8 (IL-8) at 48 hours | 22.3 [12.88 to 39.23] | 14.6 [9.34 to 22.79]
  CXCL-8 (IL-8) at 72 hours: number analyzed (Participants) | 12 | 17
  CXCL-8 (IL-8) at 72 hours | 14.5 [8.95 to 23.82] | 14.1 [9.79 to 20.39]
  CXCL-8 (IL-8) at 120 hours: number analyzed (Participants) | 10 | 11
  CXCL-8 (IL-8) at 120 hours | 10.0 [6.11 to 16.82] | 11.8 [7.73 to 17.84]
  IL-6 at 12 hours: number analyzed (Participants) | 14 | 16
  IL-6 at 12 hours | 316.2 [202.69 to 494.51] | 313.9 [210.72 to 450.05]
  IL-6 at 24 hours: number analyzed (Participants) | 14 | 17
  IL-6 at 24 hours | 317.9 [167.09 to 610.13] | 231.6 [130.64 to 402.86]
  IL-6 at 48 hours: number analyzed (Participants) | 11 | 15
  IL-6 at 48 hours | 310.5 [157.27 to 642.58] | 159.8 [88.52 to 293.27]
  IL-6 at 72 hours: number analyzed (Participants) | 12 | 16
  IL-6 at 72 hours | 249.9 [103.53 to 625.68] | 180.7 [87.50 to 383.61]
  IL-6 at 120 hours: number analyzed (Participants) | 10 | 10
  IL-6 at 120 hours | 142.2 [55.63 to 397.01] | 66.2 [27.37 to 156.20]
  RAGE at 12 hours: number analyzed (Participants) | 14 | 17
  RAGE at 12 hours | 3746 [2994.0 to 4706.5] | 3461 [2886.2 to 4174.2]
  RAGE at 24 hours: number analyzed (Participants) | 14 | 18
  RAGE at 24 hours | 3059 [2280.9 to 4094.4] | 3054 [2389.0 to 3868.3]
  RAGE at 48 hours: number analyzed (Participants) | 11 | 16
  RAGE at 48 hours | 2531 [1563.5 to 4073.7] | 2480 [1689.0 to 3665.5]
  RAGE at 72 hours: number analyzed (Participants) | 11 | 16
  RAGE at 72 hours | 1936 [1149.2 to 3357.7] | 1755 [1140.0 to 2710.0]
  RAGE at 120 hours: number analyzed (Participants) | 10 | 12
  RAGE at 120 hours | 1252 [724.6 to 2267.7] | 1292 [779.5 to 2135.8]
  MPO at 12 hours: number analyzed (Participants) | 14 | 17
  MPO at 12 hours | 60161.0 [47838.62 to 75187.43] | 65791.2 [54185.59 to 79462.44]
  MPO at 24 hours: number analyzed (Participants) | 14 | 17
  MPO at 24 hours | 55141.5 [43437.70 to 69808.68] | 69059.0 [56628.25 to 84474.33]
  MPO at 48 hours: number analyzed (Participants) | 9 | 14
  MPO at 48 hours | 58717.0 [44179.56 to 77559.82] | 73790.1 [58940.31 to 92336.24]
  MPO at 72 hours: number analyzed (Participants) | 12 | 17
  MPO at 72 hours | 42521.0 [28395.50 to 63099.18] | 60700.1 [43874.43 to 84341.04]
  MPO at 120 hours: number analyzed (Participants) | 10 | 12
  MPO at 120 hours | 32313.1 [18853.46 to 55926.54] | 47835.2 [29762.70 to 78945.65]
  Angiopoietin-2 at 12 hours: number analyzed (Participants) | 14 | 17
  Angiopoietin-2 at 12 hours | 10816.2 [8386.58 to 13875.32] | 8981.1 [7262.21 to 11069.75]
  Angiopoietin-2 at 24 hours: number analyzed (Participants) | 14 | 18
  Angiopoietin-2 at 24 hours | 9127.2 [7112.04 to 11768.48] | 8973.9 [7307.81 to 11015.23]
  Angiopoietin-2 at 48 hours: number analyzed (Participants) | 11 | 16
  Angiopoietin-2 at 48 hours | 9546.3 [7228.39 to 12627.37] | 9043.3 [7276.97 to 11310.46]
  Angiopoietin-2 at 72 hours: number analyzed (Participants) | 11 | 16
  Angiopoietin-2 at 72 hours | 8859.1 [6597.11 to 11878.90] | 7773.7 [6130.32 to 9864.61]
  Angiopoietin-2 at 120 hours: number analyzed (Participants) | 10 | 12
  Angiopoietin-2 at 120 hours | 7047.7 [4907.43 to 10244.03] | 6604.4 [4861.69 to 9194.97]
  Renin at 72 hours: number analyzed (Participants) | 15 | 16
  Renin at 72 hours | 19.95 [10.037 to 39.134] | 13.60 [7.093 to 26.212]
  Aldosterone at 72 hours: number analyzed (Participants) | 7 | 11
  Aldosterone at 72 hours | 36.8 [7.46 to 179.86] | 19.5 [7.45 to 50.56]
Statistical Analysis 1: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); CXCL-8 (IL-8), Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 12 hours; Test type: Superiority or Other; p = 0.06828, Bayesian repeated measures model; Ratio of Active/Placebo = 0.88, 95% CI 2-sided [0.528 to 1.501]
Statistical Analysis 2: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); CXCL-8 (IL-8), Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24 hours; Test type: Superiority or Other; p = 0.5674, Bayesian repeated measures model; Ratio of Active/Placebo = 0.96, 95% CI 2-sided [0.570 to 1.609]
Statistical Analysis 3: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); CXCL-8 (IL-8), Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48 hours; Test type: Superiority or Other; p = 0.8855, Bayesian repeated measures model; Ratio of Active/Placebo = 0.66, 95% CI 2-sided [0.321 to 1.316]
Statistical Analysis 4: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); CXCL-8 (IL-8), Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority; p = 0.5358, Bayesian repeated measures model; Ratio of Active/Placebo = 0.97, 95% CI 2-sided [0.531 to 1.760]
Statistical Analysis 5: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); CXCL-8 (IL-8), Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 120 hours; Test type: Superiority or Other; p = 0.6990, Bayesian repeated measures model; Ratio of Active/Placebo = 1.17, 95% CI 2-sided [0.622 to 2.155]
Statistical Analysis 6: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); IL-6, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 12 hours; Test type: Superiority or Other; p = 0.5130, Bayesian repeated measures model; Ratio of Active/Placebo = 0.99, 95% CI 2-sided [0.549 to 1.721]
Statistical Analysis 7: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); IL-6, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24 hours; Test type: Superiority or Other; p = 0.7696, Bayesian repeated measures model; Ratio of Active/Placebo = 0.73, 95% CI 2-sided [0.300 to 1.731]
Statistical Analysis 8: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); IL-6, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48 hours; Test type: Superiority or Other; p = 0.9254, Bayesian repeated measures model; Ratio of Active/Placebo = 0.51, 95% CI 2-sided [0.203 to 1.289]
Statistical Analysis 9: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); IL-6, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority or Other; p = 0.7088, Bayesian repeated measures model; Ratio of Active/Placebo = 0.72, 95% CI 2-sided [0.216 to 2.419]
Statistical Analysis 10: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); IL-6, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 120 hours; Test type: Superiority or Other; p = 0.8787, Bayesian repeated measures model; Ratio of Active/Placebo = 0.47, 95% CI 2-sided [0.112 to 1.690]
Statistical Analysis 11: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); RAGE, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 12 hours; Test type: Superiority or Other; p = 0.7338, Bayesian repeated measures model; Ratio of Active/Placebo = 0.92, 95% CI 2-sided [0.714 to 1.197]
Statistical Analysis 12: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); RAGE, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24 hours; Test type: Superiority or Other; p = 0.4955, Bayesian repeated measures model; Ratio of Active/Placebo = 1.00, 95% CI 2-sided [0.703 to 1.415]
Statistical Analysis 13: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); RAGE, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48 hours; Test type: Superiority or Other; p = 0.5264, Bayesian repeated measures model; Ratio of Active/Placebo = 0.98, 95% CI 2-sided [0.541 to 1.788]
Statistical Analysis 14: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); RAGE, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority or Other; p = 0.6183, Bayesian repeated measures model; Ratio of Active/Placebo = 0.91, 95% CI 2-sided [0.454 to 1.742]
Statistical Analysis 15: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); RAGE, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 120 hours; Test type: Superiority or Other; p = 0.5291, Bayesian repeated measures model; Ratio of Active/Placebo = 1.03, 95% CI 2-sided [0.483 to 2.118]
Statistical Analysis 16: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); MPO, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 12 hours; Test type: Superiority or Other; p = 0.7400, Bayesian repeated measures model; Ratio of Active/Placebo = 1.09, 95% CI 2-sided [0.828 to 1.448]
Statistical Analysis 17: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); MPO, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24 hours; Test type: Superiority or Other; p = 0.9375, Bayesian repeated measures model; Ratio of Active/Placebo = 1.25, 95% CI 2-sided [0.937 to 1.683]
Statistical Analysis 18: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); MPO, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48 hours; Test type: Superiority or Other; p = 0.9118, Bayesian repeated measures model; Ratio of Active/Placebo = 1.26, 95% CI 2-sided [0.896 to 1.771]
Statistical Analysis 19: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); MPO, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority or Other; p = 0.9217, Bayesian repeated measures model; Ratio of Active/Placebo = 1.43, 95% CI 2-sided [0.866 to 2.382]
Statistical Analysis 20: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); MPO, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 120 hours; Test type: Superiority or Other; p = 0.8676, Bayesian repeated measures model; Ratio of Active/Placebo = 1.48, 95% CI 2-sided [0.730 to 3.064]
Statistical Analysis 21: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Angiopoietin-2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 12 hours; Test type: Superiority or Other; p = 0.8835, Bayesian repeated measures model; Ratio of Active/Placebo = 0.83, 95% CI 2-sided [0.609 to 1.135]
Statistical Analysis 22: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Angiopoietin-2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24 hours; Test type: Superiority or Other; p = 0.5446, Bayesian repeated measures model; Ratio of Active/Placebo = 0.98, 95% CI 2-sided [0.723 to 1.330]
Statistical Analysis 23: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Angiopoietin-2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48 hours; Test type: Superiority or Other; p = 0.6267, Bayesian repeated measures model; Ratio of Active/Placebo = 0.95, 95% CI 2-sided [0.679 to 1.333]
Statistical Analysis 24: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Angiopoietin-2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority or Other; p = 0.7668, Bayesian repeated measures model; Ratio of Active/Placebo = 0.88, 95% CI 2-sided [0.612 to 1.260]
Statistical Analysis 25: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Angiopoietin-2, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 120 hours; Test type: Superiority or Other; p = 0.6100, Bayesian repeated measures model; Ratio of Active/Placebo = 0.94, 95% CI 2-sided [0.588 to 1.509]
Statistical Analysis 26: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Renin, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority or Other; p = 0.8159, Bayesian repeated measures model; Ratio of Active/Placebo = 0.68, 95% CI 2-sided [0.291 to 1.623]
Statistical Analysis 27: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); Aldosterone, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority or Other; p = 0.7988, Bayesian repeated measures model; Ratio of Active/Placebo = 0.53, 95% CI 2-sided [0.106 to 2.657]

30. Secondary Outcome: Biomarker Analysis for Serum Inflammatory Biomarker C-reactive Protein (CRP) Upto Day 5 (Part B)
Description: Serum inflammatory biomarker included CRP. Blood samples for biomarker analyses were collected 12 hours, 24 hours, 48 hours, 72 hours and 120 hours upto Day 5. Data has been presented for median along with the 95% credible interval.
Time Frame: 12 hours, 24 hours, 48 hours, 72 hours and 120 hours upto Day 5
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Median (95% Confidence Interval); unit: milligrams per deciliter
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
milligrams per deciliter
  CRP at 12 hours: number analyzed (Participants) | 14 | 17
  CRP at 12 hours | 12.99 [8.457 to 19.919] | 14.58 [10.196 to 20.872]
  CRP at 24 hours: number analyzed (Participants) | 14 | 18
  CRP at 24 hours | 11.26 [8.261 to 15.241] | 14.68 [11.357 to 18.895]
  CRP at 48 hours: number analyzed (Participants) | 11 | 16
  CRP at 48 hours | 11.19 [7.716 to 16.556] | 13.71 [9.846 to 19.529]
  CRP at 72 hours: number analyzed (Participants) | 12 | 17
  CRP at 72 hours | 9.96 [5.783 to 17.406] | 8.96 [5.510 to 14.764]
  CRP at 120 hours: number analyzed (Participants) | 10 | 11
  CRP at 120 hours | 6.81 [3.394 to 14.053] | 8.78 [4.503 to 17.514]
Statistical Analysis 1: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); CRP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 12 hours; Test type: Superiority or Other; p = 0.6536, Bayesian repeated measures model; Ratio of Active/Placebo = 1.12, 95% CI 2-sided [0.626 to 2.024]
Statistical Analysis 2: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); CRP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24 hours; Test type: Superiority or Other; p = 0.9066, Bayesian repeated measures model; Ratio of Active/Placebo = 1.30, 95% CI 2-sided [0.876 to 1.955]
Statistical Analysis 3: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); CRP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48 hours; Test type: Superiority or Other; p = 0.7859, Bayesian repeated measures model; Ratio of Active/Placebo = 1.23, 95% CI 2-sided [0.723 to 2.066]
Statistical Analysis 4: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); CRP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority or Other; p = 0.6058, Bayesian repeated measures model; Ratio of Active/Placebo = 0.90, 95% CI 2-sided [0.413 to 1.963]
Statistical Analysis 5: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); CRP, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority or Other; p = 0.6921, Ratio of Active/Placebo; Ratio of Active/Placebo = 1.29, 95% CI 2-sided [0.456 to 3.632]

31. Secondary Outcome: Biomarker Analysis for Markers of Lung Epithelial Cell Injury Clara Cell Protein 16 [CCP16]) and Surfactant Protein D [SP-D] Upto Day 5 (Part B)
Description: Markers of lung epithelial cell injury included CCP16 and SP-D. Blood samples for biomarker analyses were collected 12 hours, 24 hours, 48 hours, 72 hours and 120 hours upto Day 5. Data has been presented for median along with the 95% credible interval.
Time Frame: 12 hours, 24 hours, 48 hours, 72 hours and 120 hours upto Day 5
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Median (95% Confidence Interval); unit: nanograms per milliliter
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
nanograms per milliliter
  CCP-16 at 12 hours: number analyzed (Participants) | 14 | 17
  CCP-16 at 12 hours | 9.24 [7.771 to 10.908] | 8.45 [7.265 to 9.832]
  CCP-16 at 24 hours: number analyzed (Participants) | 13 | 17
  CCP-16 at 24 hours | 9.18 [7.525 to 11.222] | 9.25 [7.795 to 11.116]
  CCP-16 at 48 hours: number analyzed (Participants) | 11 | 14
  CCP-16 at 48 hours | 9.91 [6.784 to 14.461] | 11.04 [7.909 to 15.554]
  CCP-16 at 72 hours: number analyzed (Participants) | 12 | 17
  CCP-16 at 72 hours | 9.04 [7.232 to 11.367] | 8.94 [7.439 to 10.795]
  CCP-16 at 120 hours: number analyzed (Participants) | 10 | 12
  CCP-16 at 120 hours | 8.94 [7.067 to 11.382] | 7.22 [5.714 to 9.115]
  SP-D at 12 hours: number analyzed (Participants) | 14 | 18
  SP-D at 12 hours | 304.71 [260.328 to 357.195] | 384.58 [338.077 to 438.326]
  SP-D at 24 hours: number analyzed (Participants) | 13 | 17
  SP-D at 24 hours | 348.51 [287.860 to 421.778] | 442.35 [377.745 to 518.505]
  SP-D at 48 hours: number analyzed (Participants) | 11 | 15
  SP-D at 48 hours | 307.00 [230.616 to 405.042] | 494.70 [391.578 to 628.342]
  SP-D at 72 hours: number analyzed (Participants) | 12 | 16
  SP-D at 72 hours | 281.79 [199.927 to 398.960] | 465.15 [344.549 to 625.405]
  SP-D at 120 hours: number analyzed (Participants) | 10 | 11
  SP-D at 120 hours | 229.94 [149.118 to 349.968] | 350.31 [238.257 to 518.552]
Statistical Analysis 1: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); CCP-16, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 12 hours; Test type: Superiority or Other; p = 0.7934, Bayesian repeated measures model; Ratio of Active/Placebo = 0.92, 95% CI 2-sided [0.737 to 1.140]
Statistical Analysis 2: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); CCP-16, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24 hours; Test type: Superiority or Other; p = 0.5205, Bayesian repeated measures model; Ratio of Active/Placebo = 1.01, 95% CI 2-sided [0.782 to 1.317]
Statistical Analysis 3: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); CCP-16, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48 hours; Test type: Superiority or Other; p = 0.6682, Bayesian repeated measures model; Ratio of Active/Placebo = 1.12, 95% CI 2-sided [0.673 to 1.865]
Statistical Analysis 4: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); CCP-16, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority or Other; p = 0.5304, Bayesian repeated measures model; Ratio of Active/Placebo = 0.99, 95% CI 2-sided [0.744 to 1.315]
Statistical Analysis 5: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); CCP-16, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 120 hours; Test type: Superiority or Other; p = 0.9078, Bayesian repeated measures model; Ratio of Active/Placebo = 0.81, 95% CI 2-sided [0.582 to 1.112]
Statistical Analysis 6: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); SP-D, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 12 hours; Test type: Superiority or Other; p = 0.9907, Bayesian repeated measures model; Ratio of Active/Placebo = 1.26, 95% CI 2-sided [1.042 to 1.526]
Statistical Analysis 7: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); SP-D, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 24 hours; Test type: Superiority or Other; p = 0.9973, Bayesian repeated measures model; Ratio of Active/Placebo = 1.27, 95% CI 2-sided [1.005 to 1.606]
Statistical Analysis 8: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); SP-D, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 48 hours; Test type: Superiority or Other; p = 0.9954, Bayesian repeated measures model; Ratio of Active/Placebo = 1.61, 95% CI 2-sided [1.130 to 2.331]
Statistical Analysis 9: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); SP-D, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 72 hours; Test type: Superiority or Other; p = 0.9830, Bayesian repeated measures model; Ratio of Active/Placebo = 1.65, 95% CI 2-sided [1.045 to 2.588]
Statistical Analysis 10: Comparison: Part B (Placebo BID) vs Part B (GSK2586881 BID); SP-D, Part B (Placebo BID) Vs Part B (GSK2586881 BID) at 120 hours; Test type: Superiority or Other; p = 0.9312, Bayesian repeated measures model; Ratio of Active/Placebo = 1.52, 95% CI 2-sided [0.867 to 2.737]

32. Secondary Outcome: Immunogenicity Assessment With Respect to Anti-Acetychollinesterase2 (ACE2) Binding Antibodies at Follow-up Day 14 and Follow-up Day 28 (Part A)
Description: Blood samples for immunogenicity analysis were collected at follow-up (Day 14) and follow-up (Day 28). Antibodies to GSK2586881 were measured using a validated electrochemiluminescence bridging assay. All pre-dose and post-dose samples were first tested for Anti-ACE2 binding antibodies by screening and confirmation assay steps. The post-dose samples tested positive for anti-ACE2 binding antibodies were further characterized for anti-ACE2 neutralizing antibodies. Testing was conducted using a tiered approach; samples were first tested in a screening assay, only samples found positive in this assay were tested in the confirmation assay.
Time Frame: Follow-up (Day 14) and follow-up (Day 28)
Population: The All Subjects - Part A Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Part A
Number analyzed (Participants) | 5
Participants
  Day 14, Screening positive Confirmed negative: number analyzed (Participants) | 2
  Day 14, Screening positive Confirmed negative | 1
  Day 14, Screening positive and Confirmed positive: number analyzed (Participants) | 2
  Day 14, Screening positive and Confirmed positive | 0
  Day 14, Screening negative: number analyzed (Participants) | 2
  Day 14, Screening negative | 1
  Day 28, Screening positive Confirmed negative: number analyzed (Participants) | 1
  Day 28, Screening positive Confirmed negative | 0
  Day 28, Screening positive and Confirmed positive: number analyzed (Participants) | 1
  Day 28, Screening positive and Confirmed positive | NA — As there were no positive values at screening assay.
  Row 6, Screening negative: number analyzed (Participants) | 1
  Row 6, Screening negative | 1

33. Secondary Outcome: Immunogenicity Assessment With Respect to Anti-ACE2 Binding Antibodies at Follow-up Day 14 and Follow-up Day 28 (Part B)
Description: as for outcome 32
Time Frame: Follow-up (Day 14 )and follow-up (Day 28)
Population: The All Subjects - Part B Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Part B (Placebo BID) | Part B (GSK2586881 BID)
Number analyzed (Participants) | 20 | 19
Participants
  Day 14, Screening positive Confirmed negative: number analyzed (Participants) | 9 | 13
  Day 14, Screening positive Confirmed negative | 1 | 0
  Day 14, Screening positive and Confirmed positive: number analyzed (Participants) | 9 | 13
  Day 14, Screening positive and Confirmed positive | 0 | NA — As there were no positive values at screening assay.
  Day 14, Screening negative: number analyzed (Participants) | 9 | 13
  Day 14, Screening negative | 8 | 13
  Day 28, Screening positive Confirmed negative: number analyzed (Participants) | 10 | 11
  Day 28, Screening positive Confirmed negative | 0 | 0
  Day 28, Screening positive and Confirmed positive: number analyzed (Participants) | 10 | 11
  Day 28, Screening positive and Confirmed positive | NA — As there were no positive values at screening assay. | NA — As there were no positive values at screening assay.
  Day 28, Screening negative: number analyzed (Participants) | 10 | 11
  Day 28, Screening negative | 10 | 11

ADVERSE EVENTS:
Time Frame: Upto follow-up Day 7.
Description: The All subjects population was used for analysis.
Arm/Group | Part A | Part B (Placebo BID) | Part B (GSK2586881 BID)
All-Cause Mortality (participants affected / at risk) | 3/5 | 2/20 | 1/19
Serious Adverse Events (participants affected / at risk) | 3/5 | 4/20 | 3/19
Other Adverse Events (participants affected / at risk) | 5/5 | 14/20 | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (N=5) | Part B (Placebo BID) (N=20) | Part B (GSK2586881 BID) (N=19)
Influenza (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 1 | 0
Graft versus host disease (Immune system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Empyema (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Bronchial anastomosis complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (N=5) | Part B (Placebo BID) (N=20) | Part B (GSK2586881 BID) (N=19)
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Generalised oedema (General disorders) | 1 | 3 | 3
Injection site haemorrhage (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 6 | 3
Blood calcium decreased (Investigations) | 1 | 0 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 1 | 0 | 0
Blood sodium increased (Investigations) | 1 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 4 | 5
Insomnia (Psychiatric disorders) | 1 | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 5 | 6
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Food intolerance (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 3 | 4
Confusional state (Psychiatric disorders) | 0 | 1 | 1
Hallucination (Psychiatric disorders) | 0 | 1 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 5
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 3
Asthenia (General disorders) | 0 | 1 | 2
Peripheral swelling (General disorders) | 0 | 0 | 2
Catheter site haemorrhage (General disorders) | 0 | 1 | 0
Drug withdrawal syndrome (General disorders) | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 1
Local swelling (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2
Haemoglobin decreased (Investigations) | 0 | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0
Blood pH increased (Investigations) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0
Blood sodium increased (Investigations) | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Platelet count increased (Investigations) | 0 | 0 | 1
Respiratory rate increased (Investigations) | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2
Candiduria (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 0 | 1
Nasal herpes (Infections and infestations) | 0 | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cyanosis (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Penis injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Scrotal erythema (Reproductive system and breast disorders) | 0 | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 1 | 0
Endotracheal intubation (Surgical and medical procedures) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.